CLINICAL TRIAL: NCT04089566
Title: Escalating Dose and Randomized, Controlled Study of Nusinersen (BIIB058) in Participants With Spinal Muscular Atrophy
Brief Title: Study of Nusinersen (BIIB058) in Participants With Spinal Muscular Atrophy
Acronym: DEVOTE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 232SM203; 2019-002663-10 (EudraCT Number)
Record Dates: First submitted 2019-09-11; First posted 2019-09-13 (Actual); Results first posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Muscular Atrophy, Spinal
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — nusinersen

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 28/28 Milligram (mg) Safety Group (Experimental): Part A: Participants with later-onset SMA will receive loading doses of 28 mg of nusinersen intrathecally on Days 1, 15 and 29 followed by maintenance doses of 28 mg on Days 149 and 269.
  Interventions: Drug: Nusinersen
- 12/12 mg Active Control Group (Active Comparator): Part B: Participants with infantile- or later-onset SMA will receive loading doses of 12 mg of nusinersen intrathecally on Days 1, 15, 29, and 64 followed by maintenance doses of 12 mg on Days 183 and 279. Sham procedure will be administered on Day 135.
  Interventions: Drug: Nusinersen
- 50/28 mg Active Treatment Group (Experimental): Part B: Participants with infantile- or later-onset SMA will receive loading doses of 50 mg of nusinersen intrathecally on Days 1 and 15 followed by maintenance doses of 28 mg on Days 135 and 279. Sham procedure will be administered on Days 29, 64 and 183.
  Interventions: Drug: Nusinersen
- 12/50/28 mg Titration Group (Experimental): Part C: Participants who have been receiving the approved dose of 12 mg for at least 1 year prior to entry, will receive a single bolus dose of 50 mg of nusinersen intrathecally on Day 1 (4 months after their most recent maintenance dose of 12 mg) followed by maintenance doses of 28 mg on Days 121 and 241.
  Interventions: Drug: Nusinersen

INTERVENTIONS:
Drug: Nusinersen — Administered as specified in the treatment arm
  Other Names: BIIB058

SUMMARY:
The primary objectives of this study are to examine the clinical efficacy of nusinersen administered intrathecally at higher doses to participants with spinal muscular atrophy (SMA), as measured by change in Children's Hospital of Philadelphia-Infant Test of Neuromuscular Disorders (CHOP-INTEND) total score (Part B); to examine the safety and tolerability of nusinersen administered intrathecally at higher doses to participants with SMA (Parts A and C).

The secondary objectives of this study are to examine the clinical efficacy of nusinersen administered intrathecally at higher doses to participants with SMA (Parts A, B and C); to examine the effect of nusinersen administered intrathecally at higher doses to participants with SMA (Parts A and C); to examine the safety and tolerability of nusinersen administered intrathecally at higher doses to participants with SMA, to examine the effect of nusinersen administered intrathecally at higher doses compared to the currently approved dose in participants with SMA (Part B).

ELIGIBILITY:
Key Inclusion Criteria:

Part A, B and C:

- Genetic documentation of 5q SMA (homozygous gene deletion, mutation, or compound heterozygote)

Part A:

* Onset of clinical signs and symptoms consistent with SMA at > 6 months (> 180 days) of age (i.e., later-onset SMA)
* Age 2 to ≤ 15 years, inclusive, at the time of informed consent

Part B:

* Participants with SMA symptom onset ≤ 6 months (≤ 180 days) of age (infantile onset) should have age > 1 week to ≤ 7 months (≤ 210 days) at the time of informed consent
* Participants with SMA symptom onset > 6 months (> 180 days) of age (later onset):

  * Age 2 to < 10 years at the time of informed consent
  * Can sit independently but has never had the ability to walk independently
  * HFMSE score ≥ 10 and ≤ 54 at Screening

Part C:

- Currently on nusinersen treatment at the time of Screening, with the first dose being at least 1 year prior to Screening

Part C Cohort 1:

- Participants of any age (individuals ≥18 years of age at Screening must be ambulatory)

Part C Cohort 2:

* Participants ≥18 years of age at Screening (can be ambulatory or nonambulatory)
* HFMSE total score ≥4 points at Screening
* RULM entry item A score ≥3 points at Screening

Key Exclusion Criteria:

Part A, B and C:

* Presence of an untreated or inadequately treated active infection requiring systemic antiviral or antimicrobial therapy at any time during the Screening period
* Presence of an implanted shunt for the drainage of cerebrospinal fluid (CSF) or of an implanted central nervous system (CNS) catheter
* Hospitalization for surgery, pulmonary event, or nutritional support within 2 months prior to Screening or planned within 12 months after the participant's first dose

Part A:

* Respiratory insufficiency, defined by the medical necessity for invasive or noninvasive ventilation for > 6 hours during a 24-hour period, at Screening
* Medical necessity for a gastric feeding tube
* Treatment with an investigational drug given for the treatment of SMA, biological agent, or device within 30 days or 5 half-lives of the agent, whichever is longer, prior to Screening or anytime during the study; any prior or current treatment with any survival motor neuron-2 gene (SMN2)-splicing modifier or gene therapy; or prior antisense oligonucleotide treatment, or cell transplantation

Part B:

* Treatment with an investigational drug including but not limited to the treatment of SMA, biological agent, or device within 30 days or 5 half-lives of the agent, whichever is longer, prior to Screening or anytime during the study; any prior or current treatment with any SMN2-splicing modifier or gene therapy; or prior antisense oligonucleotide treatment, or cell transplantation
* Participants with SMA symptom onset > 6 months (> 180 days) of age (later onset):

  * Respiratory insufficiency, defined by the medical necessity for invasive or noninvasive ventilation for > 6 hours during a 24-hour period, at Screening
  * Medical necessity for a gastric feeding tube
* Participants with SMA symptom onset ≤ 6 months (≤ 180 days) of age (infantile onset): Signs or symptoms of SMA present at birth or within the first week after birth

Part C:

* Concurrent or previous participation and/or administration of nusinersen in another clinical study
* Concomitant or previous administration of any SMN2-splicing modifier (excluding nusinersen) or gene therapy, either in a clinical study or as part of medical care.
* Concurrent or previous participation in any interventional investigational study for any other drug or device within 30 days or 5 half-lives of the agent, whichever is longer, prior to Screening

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2020-03-26 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (45):
- United States (7):
  - Stanford Hospital and Clinics, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - The University of Texas Southwestern Medical Center, Dallas, Texas
- Brazil (3):
  - HC-UFMG - Hospital das Clinicas da Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital das Clínicas da Faculdade de Medicina da USP, São Paulo, São Paulo
- London Health Sciences Centre (LHSC) - Children's Hospital, London, Ontario, Canada
- Chile (3):
  - Hospital Luis Calvo Mackenna, Santiago
  - Clinica Las Condes, Santiago
  - Clinica MEDS La Dehesa, Santiago
- China (4):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - The Children's Hospital of Zhejiang University school of Med_Hangzhou, Hangzhou, Binjiang
  - Guangzhou Woman and Children's Medical Center, Guangzhou, Guangzhou
  - Xiangya Hospital, Central South University, Changsha, Hu'nan
- Colombia (2):
  - Hospital Universitario San Ignacio, Bogotá
  - Fundacion Hospitalaria San Vicente de Paul, Medellín
- Tallinn Children's Hospital, Tallinn, Estonia
- Germany (2):
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitaetsklinikum Giessen und Marburg GmbH, Giessen, Hesse
- Hungary (2):
  - Semmelweis Egyetem, Budapest
  - Magyarorszagi Reformatus Egyhaz Bethesda Gyermekkorhaz, Budapest
- Italy (2):
  - Fondazione Serena Onlus - Centro Clinico Nemo, Milan
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
- Japan (3):
  - Kurume University Hospital, Kurume-shi, Fukuoka
  - Hyogo College of Medicine Hospital, Nishinomiya-shi, Hyōgo
  - Tokyo Women's Medical University Hospital, Shinjuku-ku, Tokyo-To
- Saint George University Hospital Medical Center, Beirut, Lebanon
- Mexico (3):
  - Antiguo Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara, Jalisco
  - Instituto Nacional de Pediatria, Mexico City, Mexico City
  - Hospital Infantil de Mexico Federico Gomez, Mexico City, Mexico City
- Instytut Pomnik - Centrum Zdrowia Dziecka, Warsaw, Poland
- Russia (2):
  - Russian Children Neuromuscular Center of Veltischev, Moskva
  - Regional Pediatric Clinical Hospital #1, Yekaterinburg
- Saudi Arabia (3):
  - King Fahad Specialist Hospital, Dammam
  - National Guard Health Affairs: King Abdulaziz Medical City, Jeddah
  - King Faisal Specialist Hospital & Research Center, Riyadh
- Spain (3):
  - Hospital Sant Joan de Deu, Esplugues Del Llobregat, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitari i Politecnic La Fe, Valencia
- Taiwan (2):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

REFERENCES:
- [Derived] Finkel RS, Crawford TO, Mercuri E, Sumner CJ, Garcia Romero MDM, Day JW, Montes J, Sun P, Tichler B, Paradis AD, Boesch E, Inra J, Littauer R, Sohn J, Monine M, Gambino G, Foster R, Farewell R, Fradette S. High-dose nusinersen for spinal muscular atrophy: a phase 3 randomized trial. Nat Med. 2026 Feb 3. doi: 10.1038/s41591-025-04193-6. Online ahead of print. PMID 41634391
- [Derived] Wang X, Zheng Y, Lu J, Li X, Chen S, Xue Y, Hu S, Peng G, Zhang F, Zhao X, Liu Y, Fan Y, Zhou H, Liang C, Liu L, He L, Zhang J, Shi W, Tian J, Han M, Xu K. Musculoskeletal deformities in children with spinal muscular atrophy: a multicenter cross-sectional study with longitudinal follow-up. Ann Phys Rehabil Med. 2026 Jan 8;69(3):102080. doi: 10.1016/j.rehab.2025.102080. Online ahead of print. PMID 41512690
- [Derived] Finkel RS, Ryan MM, Pascual Pascual SI, Day JW, Mercuri E, De Vivo DC, Foster R, Montes J, Gurgel-Giannetti J, MacCannell D, Berger Z. Scientific rationale for a higher dose of nusinersen. Ann Clin Transl Neurol. 2022 Jun;9(6):819-829. doi: 10.1002/acn3.51562. Epub 2022 May 13. PMID 35567345
- See also: SMA Europe — http://www.sma-europe.eu/
- See also: CureSMA — http://www.curesma.org/
- See also: Muscular Dystrophy Association — http://www.mda.org/disease/spinal-muscular-atrophy
- See also: Study website - US patients only — https://www.biogentriallink.com/en-us/home.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at the investigative sites in the United States, Brazil, Canada, Chile, China, Colombia, Estonia, Germany, Hungary, Italy, Japan, Lebanon, Mexico, Poland, Russia, Saudi Arabia, Spain, and Taiwan.
Pre-assignment Details: A total of 145 participants diagnosed with spinal muscular atrophy (SMA) were enrolled in the 3-parts (Parts A, B, and C). Of which, 117 of participants completed the study.
Groups:
- Part A: 28/28 Milligrams (mg) Nusinersen: Participants with later-onset SMA received 3 loading doses of 28 mg of nusinersen, intrathecally (IT), on Days 1, 15 and 29 followed by 2 maintenance doses of 28 mg on Days 149 and 269.
- Part B: Infantile-Onset SMA: 12/12 mg Nusinersen: Participants with infantile-onset SMA in the control group received 4 loading doses of 12 mg of nusinersen, IT, on Days 1, 15, 29, and 64 followed by 2 maintenance doses of 12 mg on Days 183 and 279. Sham procedure was administered on Day 135.
- Part B: Infantile-Onset SMA: 50/28 mg Nusinersen: Participants with infantile-onset SMA received 2 loading doses of 50 mg of nusinersen, IT, on Days 1 and 15 followed by 2 maintenance doses of 28 mg on Days 135 and 279. Sham procedure was administered on Days 29, 64 and 183.
- Part B: Later-Onset SMA: 12/12 mg Nusinersen: Participants with later-onset SMA in the control group received 4 loading doses of 12 mg of nusinersen, IT, on Days 1, 15, 29, and 64 followed by 2 maintenance doses of 12 mg on Days 183 and 279. Sham procedure was administered on Day 135.
- Part B: Later-Onset SMA: 50/28 mg Nusinersen: Participants with later-onset SMA received 2 loading doses of 50 mg of nusinersen, IT, on Days 1 and 15 followed by 2 maintenance doses of 28 mg on Days 135 and 279. Sham procedure was administered on Days 29, 64 and 183.
- Part C: 50/28 mg Nusinersen: Participants with infantile and later-onset SMA who had been receiving the approved dose of 12 mg for at least 1 year prior to entry, received a single bolus dose of 50 mg of nusinersen, IT, on Day 1 (4 months after their most recent maintenance dose of 12 mg) followed by 2 maintenance doses of 28 mg on Days 121 and 241.
Period: Overall Study
Arm/Group | Part A: 28/28 Milligrams (mg) Nusinersen | Part B: Infantile-Onset SMA: 12/12 mg Nusinersen | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen | Part B: Later-Onset SMA: 12/12 mg Nusinersen | Part B: Later-Onset SMA: 50/28 mg Nusinersen | Part C: 50/28 mg Nusinersen
Started | 6 | 25 | 50 | 8 | 16 | 40
Completed | 6 | 13 | 35 | 7 | 16 | 40
Not Completed | 0 | 12 | 15 | 1 | 0 | 0
Not completed — Death | 0 | 6 | 10 | 0 | 0 | 0
Not completed — Withdrawal by Parent or Guardian | 0 | 2 | 1 | 0 | 0 | 0
Not completed — Reason not Specified | 0 | 4 | 4 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Part A: Safety set included all participants that received at least one dose of nusinersen. Part B: The intent-to-treat (ITT) set included all participants who were randomized and received at least one dose of nusinersen. Part C: ITT set included all participants who received at least one dose of nusinersen in the current study.
Groups:
- Part A: 28/28 mg Nusinersen: Participants with later-onset SMA received 3 loading doses of 28 mg of nusinersen, IT, on Days 1, 15 and 29 followed by 2 maintenance doses of 28 mg on Days 149 and 269.
- Part B: Infantile-Onset SMA: 12/12 mg Nusinersen: Participants with infantile-onset SMA in the control group received 4 loading doses of 12 mg of nusinersen IT on Days 1, 15, 29, and 64 followed by 2 maintenance doses of 12 mg on Days 183 and 279. Sham procedure was administered on Day 135.
- Part B: Infantile-Onset SMA: 50/28 mg Nusinersen: Participants with infantile-onset SMA received 2 loading doses of 50 mg of nusinersen IT on Days 1 and 15 followed by 2 maintenance doses of 28 mg on Days 135 and 279. Sham procedure was administered on Days 29, 64 and 183.
- Part B: Later-Onset SMA: 12/12 mg Nusinersen: Participants with later-onset SMA in the control group received 4 loading doses of 12 mg of nusinersen IT on Days 1, 15, 29, and 64 followed by 2 maintenance doses of 12 mg on Days 183 and 279. Sham procedure was administered on Day 135.
- Part B: Later-Onset SMA: 50/28 mg Nusinersen: Participants with later-onset SMA received 2 loading doses of 50 mg of nusinersen IT on Days 1 and 15 followed by 2 maintenance doses of 28 mg on Days 135 and 279. Sham procedure was administered on Days 29, 64 and 183.
- Part C: 50/28 mg Nusinersen: Participants with infantile and later-onset SMA who had been receiving the approved dose of 12 mg for at least 1 year prior to entry, received a single bolus dose of 50 mg of nusinersen IT on Day 1 (4 months after their most recent maintenance dose of 12 mg) followed by 2 maintenance doses of 28 mg on Days 121 and 241.
- Total: Total of all reporting groups
Arm/Group | Part A: 28/28 mg Nusinersen | Part B: Infantile-Onset SMA: 12/12 mg Nusinersen | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen | Part B: Later-Onset SMA: 12/12 mg Nusinersen | Part B: Later-Onset SMA: 50/28 mg Nusinersen | Part C: 50/28 mg Nusinersen | Total
Number analyzed (Participants) | 6 | 25 | 50 | 8 | 16 | 40 | 145
Age, Customized [Count of Participants; unit: Participants]
  Newborns (0-27 days) | 0 | 1 | 3 | 0 | 0 | 0 | 4
  Infants and toddlers (28 days - 23 months) | 0 | 24 | 47 | 0 | 0 | 0 | 71
  Children (2 - 11 years) | 5 | 0 | 0 | 8 | 16 | 10 | 39
  Adolescents (12 - 17 years) | 1 | 0 | 0 | 0 | 0 | 6 | 7
  Adults (18 - 64 years) | 0 | 0 | 0 | 0 | 0 | 23 | 23
  From 65 - 84 years | 0 | 0 | 0 | 0 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 11 | 24 | 6 | 14 | 15 | 71
  Male | 5 | 14 | 26 | 2 | 2 | 25 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 10 | 18 | 2 | 6 | 5 | 42
  Not Hispanic or Latino | 5 | 13 | 30 | 6 | 10 | 35 | 99
  Unknown or Not Reported | 0 | 2 | 2 | 0 | 0 | 0 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 2 | 0 | 0 | 0 | 2
  Asian | 2 | 4 | 10 | 2 | 5 | 7 | 30
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 1
  White | 4 | 17 | 29 | 3 | 8 | 32 | 93
  Not Reported Due to Confidentiality Regulations | 0 | 0 | 2 | 0 | 0 | 0 | 2
  Other | 0 | 4 | 7 | 3 | 2 | 1 | 17
Children's Hospital of Philadelphia-Infant Test of Neuromuscular Disorders (CHOPINTEND) Total Score [Mean (Standard Deviation); unit: Score on scale] — The CHOP-INTEND test was designed to evaluate the motor skills of infants with signiﬁcant motor weakness. It included 16 items (capturing neck, trunk, and proximal and distal limb strength), nine of which were scored 0, 1, 2, 3, or 4, ﬁve were scored as 0, 2, or 4, one was scored as 0, 1, 2, or 4, and one as 0, 2, 3, or 4 with higher scores indicating greater muscle strength and function. Total score was calculated as the sum of scores for each item. Total score ranged from 0 (worst possible score) and 64 (best possible score) Population: ITT set included all participants who received at least one dose of nusinersen. It was planned to be assessed in the infantile-SMA onset participants of Part B.
  Score on scale
    number analyzed (Participants) | 0 | 25 | 50 | 0 | 0 | 0 | 75
    (all) |  | 19.9 (9.63) | 20.9 (10.23) |  |  |  | 20.6 (9.98)

OUTCOME MEASURES:

1. Primary Outcome: Part B Infantile-onset SMA: Change From Baseline in CHOP-INTEND Total Score for 50/28mg Nusinersen Versus CS3B Matched Sham Control Group
Description: The CHOP-INTEND test was designed to evaluate the motor skills of infants with signiﬁcant motor weakness. It included 16 items (capturing neck, trunk, and proximal and distal limb strength), nine of which were scored 0, 1, 2, 3, or 4, ﬁve were scored as 0, 2, or 4, one was scored as 0, 1, 2, or 4, and one as 0, 2, 3, or 4 with higher scores indicating greater muscle strength and function. Total score was calculated as the sum of scores for each item. Total score ranged from 0 (worst possible score) and 64 (best possible score). The change from baseline to Day 183 in the CHOP-INTEND total score was compared to CS3B study (NCT02193074) sham control group using the joint-rank methodology to account for mortality.
Time Frame: Baseline, Day 183
Population: As planned, analysis was performed in the Matched sham set. Matched sham set comprised of sham control participants of the CS3B study (NCT02193074) identified by a matching algorithm and all of current study 50/28 mg participants that were included in the ITT set.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on scale
Groups:
- Part B: Infantile-Onset SMA: 50/28 mg Nusinersen: Participants with infantile-onset SMA received 2 loading doses of 50 mg of nusinersen intrathecally on Days 1 and 15 followed by 2 maintenance doses of 28 mg on Days 135 and 279. Sham procedure was administered on Days 29, 64 and 183.
- CS3B Matched Sham Control Group: Historical data of participants who received sham treatment on Days 1, 15, 29, 64, 183, and 302 in the double-blind, phase 3 study CS3B (NCT02193074), was used as control in the current study.
Arm/Group | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen | CS3B Matched Sham Control Group
Number analyzed (Participants) | 50 | 20
score on scale | 42.9 [38.7 to 47.2] | 16.9 [10.1 to 23.7]
Statistical Analysis 1: Comparison: Part B: Infantile-Onset SMA: 50/28 mg Nusinersen vs CS3B Matched Sham Control Group; Test type: Superiority — The Analysis of Covariance (ANCOVA) model used rank score as response, treatment as fixed effect and disease duration at screening, baseline Hammersmith Infant Neurological Examination (HINE) Section 2 (HINE 2), baseline CHOP INTEND total score as covariates; p < 0.0001, ANCOVA; Least square (LS) mean difference = 26.06, 95% CI 2-sided [17.941 to 34.172], Standard Error of Mean 4.141

2. Primary Outcome: Parts A and C: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any unfavorable & unintended sign (including an abnormal assessment such as an abnormal laboratory value), symptom, or disease temporally associated with use of an investigational product, whether or not related to investigational product. An SAE was any untoward medical occurrence that at any dose resulted in death, in the view of Investigator, placed participant at immediate risk of death, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, resulted in a birth defect. AE and SAEs were regarded as treatment-emergent if it was present prior to receiving first dose of nusinersen in this current study and subsequently worsened in severity or was not present prior to receiving first dose of nusinersen and subsequently appeared.
Time Frame: Part A: From the first dose of the study drug up to Day 389, Part C: From the first dose of the study drug up to Day 361
Population: Part A: Safety set included all participants who received at least one dose of nusinersen. Part C: ITT set included all participants who received at least one dose of nusinersen in the current study.
Measure: Count of Participants; unit: Participants
Groups:
- Part A: Nusinersen 28/28 mg: Participants with later-onset SMA received 3 loading doses of 28 mg of nusinersen IT on Days 1, 15 and 29 followed by 2 maintenance doses of 28 mg on Days 149 and 269.
- Part C: Nusinersen 50/28 mg: Participants with infantile and later-onset SMA who had been receiving the approved dose of 12 mg for at least 1 year prior to entry, received a single bolus dose of 50 mg of nusinersen intrathecally on Day 1 (4 months after their most recent maintenance dose of 12 mg) followed by 2 maintenance doses of 28 mg on Days 121 and 241.
Arm/Group | Part A: Nusinersen 28/28 mg | Part C: Nusinersen 50/28 mg
Number analyzed (Participants) | 6 | 40
Participants
  TEAEs | 4 | 37
  TESAEs | 1 | 6

3. Primary Outcome: Parts A and C: Number of Participants With Shifts From Baseline in Clinical Laboratory Parameters (Blood Chemistry Parameters)
Description: Blood chemistry parameters included protein, albumin, creatinine, blood urea nitrogen, bilirubin (total and direct), alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase, gamma-glutamyl transferase, glucose, calcium, phosphorus, bicarbonate, chloride, sodium, potassium, cystatin C, and creatine kinase. These parameters were flagged as low, normal, or high relative to parameter's normal range or as unknown if no result was available, by the Investigator. Here, shift to low indicates values that were normal, high or unknown at baseline and shifted to low values postbaseline. Shift to high indicates values that were normal, low or unknown at baseline and shifted to high values postbaseline. The categories with at least one participant with shift from baseline in these parameters are reported.
Time Frame: Parts A and C: Baseline up to Day 302
Population: Part A: Safety set included all participants who received at least one dose of nusinersen. Part C: ITT set included all participants who received at least one dose of nusinersen in the current study. Number analyzed 'n' indicates the number of participants evaluable for analysis of the specified parameter.
Measure: Count of Participants; unit: Participants
Groups:
- Part C: Nusinersen 50/28 mg: Participants with infantile and later-onset SMA who had been receiving the approved dose of 12 mg for at least 1 year prior to entry, received a single bolus dose of 50 mg of nusinersen, IT, on Day 1 (4 months after their most recent maintenance dose of 12 mg) followed by 2 maintenance doses of 28 mg on Days 121 and 241.
Arm/Group | Part A: Nusinersen 28/28 mg | Part C: Nusinersen 50/28 mg
Number analyzed (Participants) | 6 | 40
Participants
  Alkaline Phosphatase Shift to High: number analyzed (Participants) | 6 | 39
  Alkaline Phosphatase Shift to High | 1 | 2
  Alanine Aminotransferase Shift to High: number analyzed (Participants) | 6 | 34
  Alanine Aminotransferase Shift to High | 0 | 6
  Aspartate Aminotransferase Shift to High: number analyzed (Participants) | 6 | 37
  Aspartate Aminotransferase Shift to High | 0 | 8
  Bicarbonate Shift to Low: number analyzed (Participants) | 2 | 31
  Bicarbonate Shift to Low | 1 | 6
  Bicarbonate Shift to High: number analyzed (Participants) | 2 | 40
  Bicarbonate Shift to High | 0 | 2
  Bilirubin Shift to High | 0 | 1
  Indirect Bilirubin Shift to Low: number analyzed (Participants) | 4 | 26
  Indirect Bilirubin Shift to Low | 4 | 12
  Indirect Bilirubin Shift to High | 0 | 1
  Calcium Shift to High: number analyzed (Participants) | 6 | 39
  Calcium Shift to High | 0 | 1
  Creatine Kinase Shift to High: number analyzed (Participants) | 3 | 22
  Creatine Kinase Shift to High | 0 | 1
  Chloride Shift to Low | 0 | 1
  Creatinine Shift to Low: number analyzed (Participants) | 1 | 2
  Creatinine Shift to Low | 0 | 1
  Glucose Shift to Low: number analyzed (Participants) | 6 | 37
  Glucose Shift to Low | 0 | 3
  Glucose Shift to High: number analyzed (Participants) | 5 | 33
  Glucose Shift to High | 3 | 9
  Potassium Shift to High: number analyzed (Participants) | 6 | 39
  Potassium Shift to High | 1 | 1
  Phosphate Shift to High: number analyzed (Participants) | 5 | 36
  Phosphate Shift to High | 2 | 10
  Sodium Shift to High | 0 | 1
  Urea Nitrogen Shift to Low: number analyzed (Participants) | 6 | 39
  Urea Nitrogen Shift to Low | 0 | 1
  Urea Nitrogen Shift to High: number analyzed (Participants) | 6 | 39
  Urea Nitrogen Shift to High | 1 | 3

4. Primary Outcome: Parts A and C: Number of Participants With Shifts From Baseline in Clinical Laboratory Parameters (Hematology Parameters)
Description: Hematology parameters included complete blood cell count, with diﬀerential and platelet count, and absolute neutrophil count. These parameters were flagged as low, normal, or high relative to parameter's normal range or as unknown if no result was available, by the Investigator. Here, shift to low indicates values that were normal, high or unknown at baseline and shifted to low values postbaseline. Shift to high indicates values that were normal, low or unknown at baseline and shifted to high postbaseline values. The categories with at least one participant with shift from baseline in these parameters are reported.
Time Frame: Parts A and C: Baseline up to Day 302
Population: Part A: Safety set included all participants who received at least one dose of nusinersen. Part C: ITT set included all participants who received at least one dose of nusinersen in the current study. 'Number analysed (n)' indicates the number of participants evaluable for the specified hematology parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Nusinersen 28/28 mg | Part C: Nusinersen 50/28 mg
Number analyzed (Participants) | 6 | 40
Participants
  Basophils Shift to High: number analyzed (Participants) | 3 | 37
  Basophils Shift to High | 2 | 6
  Basophils/Leukocytes Shift to High: number analyzed (Participants) | 2 | 35
  Basophils/Leukocytes Shift to High | 2 | 6
  Eosinophils Shift to High: number analyzed (Participants) | 5 | 39
  Eosinophils Shift to High | 1 | 3
  Eosinophils/Leukocytes Shift to High: number analyzed (Participants) | 4 | 36
  Eosinophils/Leukocytes Shift to High | 3 | 9
  Hematocrit Shift to Low: number analyzed (Participants) | 5 | 40
  Hematocrit Shift to Low | 0 | 2
  Hematocrit Shift to High | 1 | 0
  Hemoglobin Shift to Low | 0 | 3
  Lymphocytes Shift to High: number analyzed (Participants) | 5 | 39
  Lymphocytes Shift to High | 0 | 1
  Lymphocytes/Leukocytes Shift to Low: number analyzed (Participants) | 6 | 39
  Lymphocytes/Leukocytes Shift to Low | 0 | 2
  Lymphocytes/Leukocytes Shift to High: number analyzed (Participants) | 6 | 36
  Lymphocytes/Leukocytes Shift to High | 0 | 3
  Monocytes Shift to Low: number analyzed (Participants) | 4 | 39
  Monocytes Shift to Low | 1 | 4
  Monocytes/Leukocytes Shift to Low: number analyzed (Participants) | 4 | 35
  Monocytes/Leukocytes Shift to Low | 3 | 2
  Monocytes/Leukocytes Shift to High | 0 | 2
  Neutrophils Shift to Low: number analyzed (Participants) | 6 | 35
  Neutrophils Shift to Low | 0 | 5
  Neutrophils Shift to High | 0 | 2
  Neutrophils/Leukocytes Shift to Low: number analyzed (Participants) | 5 | 38
  Neutrophils/Leukocytes Shift to Low | 1 | 4
  Neutrophils/Leukocytes Shift to High: number analyzed (Participants) | 6 | 39
  Neutrophils/Leukocytes Shift to High | 0 | 2
  Platelets Shift to Low: number analyzed (Participants) | 6 | 39
  Platelets Shift to Low | 0 | 1
  Platelets Shift to High | 0 | 1
  Leukocytes Shift to Low: number analyzed (Participants) | 6 | 36
  Leukocytes Shift to Low | 0 | 3
  Leukocytes Shift to High | 0 | 3

5. Primary Outcome: Parts A and C: Number of Participants With Shifts From Baseline in Urinalysis
Description: Urinalysis included assessments of urine total protein, specific gravity, pH, protein, glucose, ketones, bilirubin, blood, red blood cells (RBC), white blood cells (WBC), epithelial cells, bacteria, casts and crystals. These parameters were flagged as low, normal, or high relative to parameter's normal range or as unknown if no result was available, by the Investigator. Here, shift to low indicates values that were normal, high or unknown at baseline and shifted to low values postbaseline. Shift to high indicates values that were normal, low or unknown at baseline and shifted to high postbaseline. The categories with at least one participant with shift from baseline in these parameters are reported.
Time Frame: Parts A and C: Baseline up to Day 302
Population: Part A: Safety set included all participants who received at least one dose of nusinersen. Part C: ITT set included all participants who received at least one dose of nusinersen in the current study. 'Number analysed (n)' indicates the number of participants evaluable for the specified urinalysis parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Nusinersen 28/28 mg | Part C: Nusinersen 50/28 mg
Number analyzed (Participants) | 6 | 40
Participants
  Specific Gravity Shift to High: number analyzed (Participants) | 5 | 40
  Specific Gravity Shift to High | 2 | 1
  pH Shift to High | 0 | 2
  Protein High/positive: number analyzed (Participants) | 5 | 38
  Protein High/positive | 4 | 9
  Glucose High/positive | 0 | 2
  Ketones High/positive: number analyzed (Participants) | 5 | 36
  Ketones High/positive | 1 | 8
  Occult Blood High/positive: number analyzed (Participants) | 6 | 38
  Occult Blood High/positive | 2 | 4
  RBC High/positive: number analyzed (Participants) | 4 | 12
  RBC High/positive | 1 | 1
  WBC High/positive: number analyzed (Participants) | 2 | 23
  WBC High/positive | 0 | 2
  Epithelial Cells High/positive: number analyzed (Participants) | 1 | 4
  Epithelial Cells High/positive | 0 | 4
  Bacteria High/positive: number analyzed (Participants) | 1 | 2
  Bacteria High/positive | 1 | 2

6. Primary Outcome: Parts A and C: Number of Participants With Shifts From Baseline in Cerebrospinal Fluid (CSF) Parameters
Description: CSF parameters included cell count, total protein, and glucose. These parameters were flagged as low, normal, or high relative to parameter's normal range or as unknown if no result was available, by the Investigator. Here, shift to low indicates values that were normal, high or unknown at baseline and shifted to low values postbaseline. Shift to high indicates values that were normal, low or unknown at baseline and shifted to high values postbaseline. The categories with at least one participant with shift from baseline in these parameters are reported.
Time Frame: Part A: Baseline up to Day 269, Part C: Baseline up to Day 241
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Nusinersen 28/28 mg | Part C: Nusinersen 50/28 mg
Number analyzed (Participants) | 6 | 40
Participants
  Glucose Shift to Low: number analyzed (Participants) | 5 | 38
  Glucose Shift to Low | 1 | 2
  Glucose Shift to High: number analyzed (Participants) | 6 | 38
  Glucose Shift to High | 0 | 2
  Protein Shift to Low: number analyzed (Participants) | 6 | 39
  Protein Shift to Low | 0 | 3
  Protein Shift to High: number analyzed (Participants) | 6 | 37
  Protein Shift to High | 0 | 8
  Erythrocytes Shift to High: number analyzed (Participants) | 5 | 34
  Erythrocytes Shift to High | 2 | 8
  Leukocytes Shift to High: number analyzed (Participants) | 5 | 36
  Leukocytes Shift to High | 1 | 6

7. Primary Outcome: Parts A and C: Number of Participants With Shifts From Baseline in Electrocardiograms (ECGs)
Description: The ECGs were assessed by the investigator to be normal, abnormal and abnormal AE. The number of participants with ECG shifts from normal to each of the categorical values denoting an abnormal scan (abnormal not AE, abnormal AE) was assessed. Shift from baseline to worst post-baseline values were reported. The categories with at least one participant with shift from baseline in ECG are reported.
Time Frame: Parts A and C: Baseline up to Day 302
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Nusinersen 28/28 mg | Part C: Nusinersen 50/28 mg
Number analyzed (Participants) | 6 | 40
Participants
  Baseline: Normal; Postbaseline: Normal | 0 | 10
  Baseline: Normal; Post-baseline: Abnormal, not AE | 3 | 12
  Baseline: Abnormal, not AE; Post-baseline: Abnormal, not AE | 3 | 17
  Baseline: Unknown; Post-baseline: Abnormal, not AE | 0 | 1

8. Primary Outcome: Parts A and C: Number of Participants With Abnormalities in Vital Sign Parameters
Description: Vital sign assessment included temperature, pulse rate, systolic blood pressure, diastolic blood pressure, and respiratory rate. As pre-specified in protocol, the criteria for determining potentially clinically relevant abnormalities in vital signs included: temperature < 36.0 and > 38.0 degrees Celsius (C), pulse rate < 60 and > 100 beats per minute (bpm), systolic blood pressure [< 90, > 140 and > 160 millimeters of mercury (mmHg)], diastolic blood pressure < 50, > 90 and > 100 mmHg and respiratory rate < 12 and > 20 breaths per minute. The categories with at least one participant with clinically relevant vital sign abnormalities are reported.
Time Frame: Parts A and C: Baseline up to Day 302
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Nusinersen 28/28 mg | Part C: Nusinersen 50/28 mg
Number analyzed (Participants) | 6 | 40
Participants
  Temperature <36.0 C | 4 | 13
  Pulse rate <60 bpm | 1 | 14
  Pulse rate >100 bpm | 6 | 19
  Systolic blood pressure <90 mmHg | 4 | 13
  Systolic blood pressure >140 mmHg | 0 | 3
  Diastolic blood pressure <50 mmHg | 1 | 7
  Diastolic blood pressure >90 mmHg | 0 | 1
  Respiratory rate <12 breaths/min | 1 | 7
  Respiratory rate >20 breaths/min | 6 | 27

9. Primary Outcome: Parts A and C: Change From Baseline in Growth Parameters (Body Height)
Time Frame: Parts A and C: Baseline, Day 302
Population: Part A: Safety set included all participants who received at least one dose of nusinersen. Part C: ITT set included all participants who received at least one dose of nusinersen in the current study. 'Overall number of participants analyzed' signifies number of participants evaluable for this outcome measure at the specified time point.
Measure: Mean (Standard Deviation); unit: centimeter (cm)
Arm/Group | Part A: Nusinersen 28/28 mg | Part C: 50/28 mg Nusinersen
Number analyzed (Participants) | 2 | 32
centimeter (cm) | 7.2 (1.70) | 0.8 (3.12)

10. Primary Outcome: Part C: Change From Baseline in Growth Parameters (Head Circumference)
Description: As pre-specified in the protocol, head circumference was measured for participants with infantile-onset SMA only.
Time Frame: Baseline, Day 302
Population: ITT set included all participants who received at least one dose of nusinersen in the current study. 'Overall number of participants analyzed' signifies number of participants evaluable for this outcome measure at the specified time point.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Part C: Nusinersen 50/28 mg
Number analyzed (Participants) | 1
cm | 2.0 (NA) — Since only one participant was evaluable, standard deviation (SD) was not estimated

11. Primary Outcome: Part C: Change From Baseline in Growth Parameters (Chest Circumference)
Description: As pre-specified in protocol, chest circumference was measured for participants with infantile-onset SMA only.
Time Frame: Baseline, Day 302
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Part C: Nusinersen 50/28 mg
Number analyzed (Participants) | 1
cm | 2.5 (NA) — Since only one participant was evaluable, SD was not estimated

12. Primary Outcome: Part C: Change From Baseline in Growth Parameters (Arm Circumference)
Description: As pre-specified in the protocol, arm circumference was measured for participants with infantile-onset SMA. Here, negative change from baseline indicated reduction in arm circumference.
Time Frame: Baseline, Day 302
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Part C: Nusinersen 50/28 mg
Number analyzed (Participants) | 1
cm | -1.0 (NA) — Since only one participant was evaluable, SD was not estimated

13. Primary Outcome: Parts A and C: Change From Baseline in Growth Parameters (Ulnar Length)
Description: As pre-specified in the protocol, ulnar length was measured for participants with later-onset SMA.
Time Frame: Parts A and C: Baseline, Day 302
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Part A: Nusinersen 28/28 mg | Part C: 50/28 mg Nusinersen
Number analyzed (Participants) | 6 | 27
cm | 1.8 (1.43) | 0.0 (1.27)

14. Primary Outcome: Parts A and C: Change From Baseline in Growth Parameters (Weight for Age Percentile)
Description: World Health Organization (WHO) child growth standards (2006) was used to calculate the weight for age percentile in the infantile-onset participants while the 2000 Centers for Disease Control and Prevention (CDC) Growth Charts was used to calculate the weight for age percentile for later-onset participants. Negative change from baseline indicates low weight for age percentile.
Time Frame: Parts A and C: Baseline, Day 302
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percentile
Arm/Group | Part A: Nusinersen 28/28 mg | Part C: 50/28 mg Nusinersen
Number analyzed (Participants) | 6 | 17
percentile | 12.2 (12.84) | -2.7 (9.47)

15. Primary Outcome: Part C: Change From Baseline in Growth Parameters (Weight for Length Ratio)
Description: As pre-specified in the protocol, weight for length ratio was assessed only for the participants with infantile-onset SMA.
Time Frame: Baseline, Day 302
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Part C: 50/28 mg Nusinersen
Number analyzed (Participants) | 1
ratio | 0.005 (NA) — Since only one participant was evaluated, SD was not estimable.

16. Primary Outcome: Part C: Change From Baseline in Growth Parameters (Head-to-Chest Circumference Ratio)
Description: As pre-specified in the protocol, head to chest circumference ratio was assessed only for the participants with infantile-onset SMA.
Time Frame: Baseline, Day 302
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Part C: Nusinersen 50/28 mg
Number analyzed (Participants) | 1
ratio | 0.0 (NA) — Since only one participant was evaluable, SD was not estimated

17. Primary Outcome: Parts A and C: Number of Participants With Shifts From Baseline in Coagulation Parameters (Activated Partial Thromboplastin Time (aPTT))
Description: Activated partial thromboplastin time was evaluated to assess safety. "Shift to low" measured change in normal, high and unknown values of aPTT at baseline to low values postbaseline. "Shift to high" measured change in normal, low and unknown values of aPTT at baseline to high values postbaseline.
Time Frame: Parts A and C: Baseline up to Day 269
Population: Part A: Safety set included all participants who received at least one dose of nusinersen. Part C:ITT set included all participants who received at least one dose of nusinersen in the current study. 'Number analysed (n)' signifies number of participants evaluable for the specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Nusinersen 28/28 mg | Part C: 50/28 mg Nusinersen
Number analyzed (Participants) | 6 | 40
Participants
  Shift to Low | 0 | 5
  Shift to High: number analyzed (Participants) | 5 | 36
  Shift to High | 0 | 1

18. Primary Outcome: Parts A and C: Number of Participants With Shifts From Baseline in Coagulation Parameters (Prothrombin Time (PT))
Description: Prothrombin time was evaluated to assess safety. "Shift to low" measured change in normal, high and unknown values of PT at baseline to low values postbaseline. "Shift to high" measured change in normal, low and unknown values of PT at baseline to high values postbaseline.
Time Frame: Parts A and C: Baseline up to Day 269
Population: Part A: Safety set included all participants who received at least one dose of nusinersen. Part C: ITT set included all participants who received at least one dose of nusinersen in the current study. 'Overall number of participants analyzed' signifies number of participants evaluable for this outcome measure. 'Number analysed (n)' signifies number of participants evaluable for the specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Nusinersen 28/28 mg | Part C: 50/28 mg Nusinersen
Number analyzed (Participants) | 6 | 34
Participants
  Shift to Low | 0 | 0
  Shift to High: number analyzed (Participants) | 6 | 32
  Shift to High | 0 | 1

19. Primary Outcome: Parts A and C: Number of Participants With Shifts From Baseline in Coagulation Parameters (International Normalized Ratio (INR))
Description: INR was evaluated to assess safety. "Shift to low" measured change in normal, high and unknown values of INR at baseline to low values postbaseline. "Shift to high" measured change in normal, low and unknown values of INR at baseline to high values postbaseline. The category with at least one participant with shift from baseline in INR ratio is reported.
Time Frame: Parts A and C: Baseline up to Day 269
Population: Part A: Safety set included all participants who received at least one dose of nusinersen. Part C: ITT set included all participants who received at least one dose of nusinersen in the current study. 'Number analysed (n)' signifies number of participants evaluable for the specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Nusinersen 28/28 mg | Part C: 50/28 mg Nusinersen
Number analyzed (Participants) | 6 | 40
Participants
  Shift to Low | 0 | 3
  Shift to High: number analyzed (Participants) | 6 | 39
  Shift to High | 0 | 0

20. Primary Outcome: Parts A and C: Change From Baseline in Urine Total Protein
Time Frame: Parts A and C: Baseline, Day 302
Population: Part A: Safety set included all participants who received at least one dose of nusinersen. Part C: ITT set included all participants who received at least one dose of nusinersen in the current study. 'Overall number of participants analyzed' signifies number of participants evaluable for this outcome measure at specified timepoint.
Measure: Mean (Standard Deviation); unit: gram per litre (g/L)
Arm/Group | Part A: Nusinersen 28/28 mg | Part C: 50/28 mg Nusinersen
Number analyzed (Participants) | 3 | 29
gram per litre (g/L) | 0.010 (0.1235) | -0.692 (3.7040)

21. Primary Outcome: Parts A and C: Number of Participants With Neurological Examination Abnormalities Reported as AEs
Description: Participants with abnormalities in neurological examinations recorded as AEs were reported.
Time Frame: Parts A and C: Baseline up to Day 302
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Nusinersen 28/28 mg | Part C: 50/28 mg Nusinersen
Number analyzed (Participants) | 6 | 40
Participants
  Vestibular Disorder | 0 | 1
  Asthenia | 0 | 1
  Gait Disturbance | 0 | 1
  Balance Disorder | 0 | 1
  Disturbance in Attention | 0 | 1
  Paraesthesia | 1 | 0

22. Primary Outcome: Parts A and C: Percentage of Participants With a Postbaseline Platelet Count Below the Lower Limit of Normal on at Least 2 Consecutive Measurements
Time Frame: Parts A and C: Baseline up to Day 302
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Part A: Nusinersen 28/28 mg | Part C: 50/28 mg Nusinersen
Number analyzed (Participants) | 6 | 40
percentage of participants | 0 | 2.5

23. Primary Outcome: Parts A and C: Percentage of Participants With a Postbaseline Corrected QT Interval Using Fridericia's Formula (QTcF) of > 500 Millisecond (Msec) and an Increase From Baseline to Any Postbaseline Timepoint in QTcF of > 60 Msec
Time Frame: Parts A and C: Baseline up to Day 302
Population: Part A: Safety set included all participants who received at least one dose of nusinersen. Part C: ITT set included all participants who received at least one dose of nusinersen in the current study. 'Overall number of participants analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Part A: Nusinersen 28/28 mg | Part C: 50/28 mg Nusinersen
Number analyzed (Participants) | 6 | 39
percentage of participants | 0 | 0

24. Secondary Outcome: Part B Infantile-onset SMA: Percentage of Hammersmith Infant Neurological Examination (HINE) Section 2 Motor Milestone Responders for Nusinersen 50/28mg Treatment Group Versus CS3B Matched Sham Control Group
Description: Section 2 of HINE was used to assess motor milestones of participants. It's composed of 8 motor milestone categories: voluntary grasp, ability to kick in supine position, head control, rolling, sitting, crawling, standing, & walking. Motor milestone responder: (i) a participant that demonstrated at least a 2-point increase in category of ability to kick or maximal score on that category or a 1-point increase in category of head control, rolling, sitting, crawling, standing, or walking, (ii) improvement in more categories than worsening, excluding category of voluntary grasp. For category of ability to kick, improvement, as defined in (i), worsening: at least a 2-point decrease or decrease to lowest possible score of no kicking. For other 6 categories, improvement: 1-point increase, worsening: at least 1-point decrease. Participants who died or withdrew from study were considered as non-responders. Difference in percentage of responders reported using Fisher's exact test.
Time Frame: Baseline, Day 183
Population: As planned, analysis was performed in the Matched sham set. Matched sham set comprised of sham control participants of CS3B study (NCT02193074) identified by a matching algorithm and all of current study 50/28 mg participants that were included in the ITT set.
Measure: Number; unit: percentage of responders
Groups:
- CS3B Matched Sham Control Group: Historical data of participants who received sham treatment, IT, on Days 1, 15, 29, 64, 183, and 302 in the double-blind, phase 3 study CS3B (NCT02193074), was used as control in the current study.
Arm/Group | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen | CS3B Matched Sham Control Group
Number analyzed (Participants) | 50 | 20
percentage of responders | 58 | 0
Statistical Analysis 1: Comparison: Part B: Infantile-Onset SMA: 50/28 mg Nusinersen vs CS3B Matched Sham Control Group; Test type: Superiority; p < 0.0001, Fisher Exact; Difference of percentages = 58, 95% CI 2-sided [39.46 to 71.81] — Exact unconditional confidence interval

25. Secondary Outcome: Part B Infantile-onset SMA: Change From Baseline in HINE Section 2 Motor Milestones Total Score for Nusinersen 50/28mg Treatment Group Versus CS3B Matched Sham Control Group
Description: Section 2 of the HINE was used to assess motor milestones of the participants. It's composed of 8 motor milestone categories: voluntary grasp, ability to kick in supine position, head control, rolling, sitting, crawling, standing, and walking. Within each category, 3 to 5 levels can be achieved. The total HINE section 2 motor milestones score was calculated as sum of each level & ranged from 0 to 26, higher score indicating improvement in motor milestones. A negative change from baseline indicates decline in motor milestones. Change from baseline in HINE section 2 motor milestones total score was compared to study CS3B (NCT02193074) matched sham control group, and was analysed using joint rank methodology.
Time Frame: Baseline, Day 183
Population: As planned, analysis was performed in the Matched sham set. Matched sham set comprised of sham control participants of CS3B study (NCT02193074) identified by a matching algorithm and all of current study 50/28 mg participants that were included in ITT set.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on scale
Arm/Group | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen | CS3B Matched Sham Control Group
Number analyzed (Participants) | 50 | 20
score on scale | 43.1 [39.0 to 47.2] | 16.5 [9.9 to 23.0]
Statistical Analysis 1: Comparison: Part B: Infantile-Onset SMA: 50/28 mg Nusinersen vs CS3B Matched Sham Control Group; Test type: Superiority; p < 0.0001, ANCOVA — ANCOVA model was used treatment as fixed effect and disease duration at screening, baseline HINE 2, baseline CHOP INTEND total score as covariates; LS mean difference = 26.67, 95% CI 2-sided [18.812 to 34.526], Standard Error of Mean 4.009

26. Secondary Outcome: Part B Infantile-onset SMA: Change From (Ratio to) Baseline in Plasma Concentration of Neurofilament Light Chain (NF-L) for 50/28mg Nusinersen Versus CS3B Matched Sham Control Group
Description: The change from baseline in the plasma concentration of NF-L was compared to the study CS3B (NCT02193074) matched sham control group. Joint rank methodology was used for the analysis to account for mortality. The change from baseline data was reported in terms of least square geometric mean ratio to baseline. Lower ratios to baseline represent greater reductions in concentrations of NF-L from baseline.
Time Frame: Baseline, Day 183
Population: as for outcome 1
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen | CS3B Matched Sham Control Group
Number analyzed (Participants) | 50 | 20
ratio | 0.06 [0.05 to 0.07] | 0.70 [0.43 to 1.12]
Statistical Analysis 1: Comparison: Part B: Infantile-Onset SMA: 50/28 mg Nusinersen vs CS3B Matched Sham Control Group; Test type: Superiority; p < 0.0001, ANCOVA — ANCOVA model was used with treatment as a fixed effect and adjusted for each participant disease duration at screening, baseline log plasma NF-L and baseline CHOP INTEND total score; LS geometric mean ratio = 0.08

27. Secondary Outcome: Part B Infantile-onset SMA: Change From Baseline in CHOP-INTEND Total Score for 50/28mg Nusinersen Versus 12/12mg Nusinersen
Description: The CHOP-INTEND test was designed to evaluate the motor skills of infants with signiﬁcant motor weakness. It included 16 items (capturing neck, trunk, and proximal and distal limb strength), nine of which were scored 0, 1, 2, 3, or 4, ﬁve were scored as 0, 2, or 4, one was scored as 0, 1, 2, or 4, and one as 0, 2, 3, or 4 with higher scores indicating greater muscle strength and function. Total score was calculated as the sum of scores for each item. Total score ranged from 0 (worst possible score) and 64 (best possible score). The change from baseline to Day 302 in the total score was analyzed using the joint-rank methodology to account for mortality.
Time Frame: Baseline, Day 302
Population: ITT set included all participants who were randomized and received at least one dose of nusinersen.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on scale
Groups:
- Part B: Infantile-Onset SMA: 12/12 mg Nusinersen: Participants with infantile-onset SMA received 4 loading doses of 12 mg of nusinersen intrathecally on Days 1, 15, 29, and 64 followed by 2 maintenance doses of 12 mg on Days 183 and 279. Sham procedure was administered on Day 135.
Arm/Group | Part B: Infantile-Onset SMA: 12/12 mg Nusinersen | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen
Number analyzed (Participants) | 25 | 50
score on scale | 37.3 [29.1 to 45.5] | 38.3 [32.7 to 44.0]
Statistical Analysis 1: Comparison: Part B: Infantile-Onset SMA: 12/12 mg Nusinersen vs Part B: Infantile-Onset SMA: 50/28 mg Nusinersen; Test type: Superiority; p = 0.8484, ANCOVA — ANCOVA model used rank score as response, treatment as fixed effect and disease duration at screening, baseline HINE 2, baseline CHOP INTEND total score as covariates; LS mean difference = 1, 95% CI 2-sided [-9.29 to 11.299], Standard Error of Mean 5.251

28. Secondary Outcome: Part B Infantile-onset SMA: Change From Baseline in HINE Section 2 Motor Milestones Total Score for 50/28mg Nusinersen Versus 12/12mg Nusinersen
Description: Section 2 of the HINE was used to assess motor milestones of the participants. It's composed of 8 motor milestone categories: voluntary grasp, ability to kick in supine position, head control, rolling, sitting, crawling, standing, and walking. Within each of these categories, participants can progress from complete absence of a motor ability (the lowest level in each category) through multiple milestones (2 to 4 levels in each category) to the highest level within the category. The total motor milestones score for HINE section was calculated as the sum of each level and ranged from 0 to a maximum score of 26, higher score indicating improvement in motor milestones.
Time Frame: Baseline, Day 302
Population: ITT set included all participants who were randomized and received at least one dose of nusinersen.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on scale
Arm/Group | Part B: Infantile-Onset SMA: 12/12 mg Nusinersen | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen
Number analyzed (Participants) | 25 | 50
score on scale | 33.9 [26.9 to 41.0] | 40.0 [35.1 to 44.9]
Statistical Analysis 1: Comparison: Part B: Infantile-Onset SMA: 12/12 mg Nusinersen vs Part B: Infantile-Onset SMA: 50/28 mg Nusinersen; Test type: Superiority; p = 0.1734, ANCOVA — [p-value comment as in outcome 27, analysis 1]; LS mean difference = 6.12, 95% CI 2-sided [-2.693 to 14.939], Standard Error of Mean 4.497

29. Secondary Outcome: Part B Infantile-onset SMA: Change From (Ratio to) Baseline in Plasma Concentration of NF-L for 50/28mg Nusinersen Versus 12/12mg Nusinersen
Description: The change from baseline in plasma concentration of NF-L was analysed using the joint rank methodology to account for mortality. The change from baseline data was reported in terms of LS geometric mean ratio to baseline. Lower ratios to baseline represent greater reductions in concentrations of NF-L from baseline.
Time Frame: Baseline, Day 64
Population: ITT set included all participants who were randomized and received at least one dose of nusinersen.
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | Part B: Infantile-Onset SMA: 12/12 mg Nusinersen | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen
Number analyzed (Participants) | 25 | 50
ratio | 0.23 [0.16 to 0.32] | 0.12 [0.09 to 0.15]
Statistical Analysis 1: Comparison: Part B: Infantile-Onset SMA: 12/12 mg Nusinersen vs Part B: Infantile-Onset SMA: 50/28 mg Nusinersen; Test type: Superiority; p = 0.002, ANCOVA — ANCOVA model was used with treatment as a fixed effect and adjustment for each participant disease duration at screening, baseline log plasma NF-L and baseline CHOP INTEND total score; LS geometric mean ratio = 0.51, 95% CI 2-sided [0.33 to 0.78]

30. Secondary Outcome: Part B Infantile-onset SMA: Time to Death or Permanent Ventilation for 50/28mg Nusinersen Versus CS3B Matched Sham Control Group
Description: Permanent ventilation was deﬁned as tracheostomy or ≥ 16 hours of ventilation/day continuously for > 21 days in absence of an acute reversible event. An independent endpoint adjudication committee (EAC) determined date at which a participant was considered to have met protocol-specified criteria of an acute reversible event. Only events that were adjudicated by the EAC as meeting the criteria for permanent ventilation or death were included in analysis. Participants who did not meet the endpoint definition were censored on the last occasion the participant was seen (either in-person visit or by telephone contact), irrespective of whether the participant has completed the full course of treatment and whether the participant has completed the study or permanently withdrawn.
Time Frame: Screening up to Day 399
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen | CS3B Matched Sham Control Group
Number analyzed (Participants) | 50 | 20
weeks | NA [39.86 to NA] — Median and confidence interval were not estimable due to low number events of permanent ventilation or death. | 19.1 [10.00 to 31.29]

31. Secondary Outcome: Part B Infantile-onset SMA: Time to Death (Overall Survival) for 50/28mg Nusinersen Versus CS3B Matched Sham Control Group
Description: Time to death was determined by an independent EAC. Time to death (overall survival) was compared to the study CS3B (NCT02193074) matched sham control group.
Time Frame: Screening up to Day 399
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- CS3B Matched Sham Control Group: Historical data of participants who received sham treatment, IT, on Days 1, 15, 29, 64, 183, and 302 in the double-blind, phase 3 study CS3B (2013-004422-29), was used as control in the current study.
Arm/Group | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen | CS3B Matched Sham Control Group
Number analyzed (Participants) | 50 | 20
weeks | NA [NA to NA] — Median and confidence interval were not estimable due to low number of events of death. | 33.6 [11.29 to NA] — Upper range 95% CI was not estimable due to low number of events of death.

32. Secondary Outcome: Part B Infantile-onset SMA: Time to Death or Permanent Ventilation for 50/28mg Nusinersen Versus 12/12mg Nusinersen
Description: Permanent ventilation was deﬁned as tracheostomy or ≥ 16 hours of ventilation/day continuously for > 21 days in the absence of an acute reversible event. An independent EAC determined the date at which a participant was considered to have met the protocol-specified criteria of an acute reversible event. Only events that were adjudicated by the EAC as meeting the protocol defined criteria for permanent ventilation or death was included in the analysis. Participants who did not meet the endpoint definition were censored on the last occasion the participant was seen (either in-person visit or by telephone contact), irrespective of whether the participant has completed the full course of treatment and whether the participant has completed the study or permanently withdrawn.
Time Frame: Screening up to Day 399
Population: ITT set included all participants who were randomized and received at least one dose of nusinersen.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Part B: Infantile-Onset SMA: 12/12 mg Nusinersen | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen
Number analyzed (Participants) | 25 | 50
weeks | 24.7 [14.43 to NA] — Upper range 95% CI was not estimable due to low number of events of permanent ventilation or death. | NA [39.86 to NA] — Median and confidence interval were not estimable due to low number of events of permanent ventilation or death.

33. Secondary Outcome: Part B Infantile-onset SMA: Time to Death (Overall Survival) for 50/28mg Nusinersen Versus 12/12mg Nusinersen
Description: Time to death was determined by an independent EAC. Participants who did not die were censored on the last occasion the participant was seen (either in-person visit or by telephone contact), irrespective of whether the participant has completed the full course of treatment and whether the participant has completed the study or permanently withdrawn.
Time Frame: Screening up to Day 399
Population: ITT set included all participants who were randomized and received at least one dose of nusinersen.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Part B: Infantile-Onset SMA: 12/12 mg Nusinersen | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen
Number analyzed (Participants) | 25 | 50
weeks | NA [24.71 to NA] — Median and confidence interval were not estimable due to low number events of death. | NA [NA to NA] — Median and confidence interval were not estimable due to low number events of death.

34. Secondary Outcome: Part B Later-onset SMA: Change From Baseline in Hammersmith Functional Motor Scale Expanded (HFMSE) Score for 50/28mg Nusinersen Versus 12/12mg Nusinersen
Description: HFMSE scale was a tool used to assess motor function in children with later-onset SMA. The original 20 item Hammersmith Functional Motor Scale was expanded to include 13 additional adapted items from the Gross Motor Function Measure to improve sensitivity for the higher functioning ambulant population. Each item is scored 0 (unable), 1 (performs with modiﬁcation or adaptation) or 2 (able) and the total score was calculated by summing the 33 items and ranged from 0 to 66 with higher scores indicating greater motor function.
Time Frame: Baseline, Day 302
Population: ITT set included all participants who were randomized and received at least one dose of nusinersen.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on scale
Groups:
- Part B: Later-Onset SMA: 12/12 mg Nusinersen: Participants with later-onset SMA received 4 loading doses of 12 mg of nusinersen intrathecally on Days 1, 15, 29, and 64 followed by 2 maintenance doses of 12 mg on Days 183 and 279. Sham procedure was administered on Day 135.
- Part B: Later-Onset SMA: 50/28 mg Nusinersen: Participants with later-onset SMA received 2 loading doses of 50 mg of nusinersen intrathecally on Days 1 and 15 followed by 2 maintenance doses of 28 mg on Days 135 and 279. Sham procedure was administered on Days 29, 64 and 183.
Arm/Group | Part B: Later-Onset SMA: 12/12 mg Nusinersen | Part B: Later-Onset SMA: 50/28 mg Nusinersen
Number analyzed (Participants) | 8 | 16
score on scale | 2.6 [0.2 to 5.1] | 3.3 [1.5 to 5.0]

35. Secondary Outcome: Part B Later-onset SMA: Change From Baseline in Revised Upper Limb Module (RULM) Score for 50/28mg Nusinersen Versus 12/12mg Nusinersen
Description: RULM test was developed to assess upper limb functional abilities. RULM test: total 20 items. First item was assessed on 7-point scale (0:No useful function to 6-Can abduct both arms simultaneously, elbows in extension in full circle until they touch above head). This first item did not contribute to total score. For remaining 19 items, 18 items were assessed on 3-point scale: 0-Unable to achieve independently; 1-Modified method but achieves goal independent of physical assistance from another person; 2-Normal -achieves goal without any assistance. One remaining item was assessed as either 0 or 1. For each item, score was collected on left & right side. Derived total score=summing scores from these 19 individual items ranging from 0-if participant fails all activities to 37-if participant achieves all activities. If, for an individual item, response was recorded for both left & right side, highest score was used in calculating total score. Higher scores=increased upper limb function.
Time Frame: Baseline, Day 302
Population: ITT set included all participants who were randomized and received at least one dose of nusinersen.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on scale
Arm/Group | Part B: Later-Onset SMA: 12/12 mg Nusinersen | Part B: Later-Onset SMA: 50/28 mg Nusinersen
Number analyzed (Participants) | 8 | 16
score on scale | 1.8 [-0.8 to 4.4] | 2.5 [0.7 to 4.2]

36. Secondary Outcome: Part B Later-onset SMA: Number of New World Health Organization (WHO) Motor Milestones Achieved Per Participant for 50/28mg Nusinersen Versus 12/12mg Nusinersen
Description: The WHO motor milestones were a set of six milestones in motor development: sitting without support, standing with assistance, hands and knees crawling, walking with assistance, standing alone and walking alone. The examiner recorded an overall rating of the participant's emotional state and then for each milestone one of the following four classiﬁcations: no (inability) - child tried but failed to perform the milestone, no (refusal) - child refused to perform despite being calm and alert, yes - child was able to perform the milestone, unable to test - could not be tested because of irritability, drowsiness or sickness. Mean of number of new milestones achieved per participant was calculated and reported in this outcome measure.
Time Frame: Baseline, Day 302
Population: ITT set included all participants who were randomized and received at least one dose of nusinersen. 'Overall number of participants analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: motor milestones per participant
Arm/Group | Part B: Later-Onset SMA: 12/12 mg Nusinersen | Part B: Later-Onset SMA: 50/28 mg Nusinersen
Number analyzed (Participants) | 7 | 16
motor milestones per participant | 0.0 (0.00) | 0.3 (1.00)

37. Secondary Outcome: Part B Later-onset SMA: Change From Baseline in Assessment of Caregiver Experience With Neuromuscular Disease (ACEND) for 50/28mg Nusinersen Versus 12/12mg Nusinersen
Description: ACEND instrument was designed to quantify caregiver impact experienced by parents/caregivers of children affected with severe neuromuscular diseases, including children with SMA. The ACEND included a total of seven domains assessing physical impact (including feeding/grooming/dressing, sitting/play, transfers, and mobility) and general caregiver impact (including time, emotion, and finance, and each domain comprised several items. The total score for each domain was calculated on a scale of 0 to 100, with a higher score indicating a decreased caregiver burden. A negative change from baseline indicates an increased caregiver burden.
Time Frame: Baseline, Day 302
Population: ITT set included all participants who were randomized and received at least one dose of nusinersen.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on scale
Arm/Group | Part B: Later-Onset SMA: 12/12 mg Nusinersen | Part B: Later-Onset SMA: 50/28 mg Nusinersen
Number analyzed (Participants) | 8 | 16
score on scale
  Feeding/Grooming/Dressing Total Score | 7.9 [-4.8 to 20.6] | 8.3 [-0.2 to 16.7]
  Sitting/Play Total Score | 10.3 [0.6 to 20.0] | 10.1 [3.6 to 16.6]
  Transfers Total Score | -0.0 [-10.9 to 10.9] | 9.9 [2.6 to 17.2]
  Mobility Total Score | 6.9 [-7.2 to 20.9] | 8.1 [-0.9 to 17.0]
  Time Total Score | -4.4 [-17.9 to 9.2] | 11.9 [2.9 to 20.9]
  Emotion Total Score | 2.6 [-8.7 to 13.9] | 2.5 [-5.0 to 10.0]
  Finance Total Score | -7.7 [-20.9 to 5.6] | 7.8 [-0.7 to 31.7]

38. Secondary Outcome: Part B Later-onset SMA: Change From Baseline in Pediatric Quality of Life Inventory™ (PedsQL) for 50/28mg Nusinersen Versus 12/12mg Nusinersen
Description: Participants were evaluated using PedsQL generic core scale & neuromuscular module. PedsQL generic core scale was used to calculate PedsQL inventory total score (PQLI), that included parent & participant's assessment on 4 dimensions: physical, emotional, social, & school functioning & psychosocial health. Each item was scored on 5-point ordinal scale (0=never to 4=almost always). PedsQL neuromuscular module (PQLN) measured HRQOL dimensions specific to with neuromuscular disorders, like SMA. Each item was scored on 5-point ordinal scale (0=never to 4=almost always). Dimensions were reversed scored & were linearly transformed to 0-100 scale (0=100, 1=75, 2=50, 3=25, 4=0) for both PQLI and PQLN, higher scores indicative of better health related quality of life. Total scale scores were calculated as sum of all items over number of items answered on all scales. If more than 50% of items/more within a dimension were missing, scale score was not computed.
Time Frame: Baseline, Day 302
Population: ITT set included all participants who were randomized and received at least one dose of nusinersen. 'Overall number of participants analyzed' signifies number of participants evaluable for this outcome measure. 'Number analysed (n)' indicates number of participants evaluable for the specified total score
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Part B: Later-Onset SMA: 12/12 mg Nusinersen | Part B: Later-Onset SMA: 50/28 mg Nusinersen
Number analyzed (Participants) | 7 | 16
score on scale
  PQLI-Total Score-Participant: number analyzed (Participants) | 4 | 12
  PQLI-Total Score-Participant | -5.1 (4.73) | 3.8 (2.61)
  PQLI-Total Score-Parent: number analyzed (Participants) | 7 | 14
  PQLI-Total Score-Parent | -9.6 (4.32) | -6.9 (2.96)
  PQLN-Total Score-Participant: number analyzed (Participants) | 4 | 12
  PQLN-Total Score-Participant | -4.8 (3.41) | 10.4 (1.91)
  PQLN-Total Score-Parent | -6.4 (4.25) | -0.7 (2.81)

39. Secondary Outcome: Part B Later-onset SMA: Change From (Ratio to) Baseline in CSF Concentration of NF-L for 50/28mg Nusinersen Versus 12/12mg Nusinersen
Description: The change from baseline data was reported in terms of geometric mean ratio to baseline. Lower ratios to baseline represent greater reductions in concentrations of NF-L from baseline.
Time Frame: Baseline, Day 279
Population: ITT set included all participants who were randomized and received at least one dose of nusinersen.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Part B: Later-Onset SMA: 12/12 mg Nusinersen | Part B: Later-Onset SMA: 50/28 mg Nusinersen
Number analyzed (Participants) | 8 | 16
ratio | 0.32 [0.23 to 0.450] | 0.33 [0.26 to 0.41]

40. Secondary Outcome: Part B Later-onset SMA: Change From (Ratio to) Baseline in Plasma Concentration of NF-L for 50/28mg Nusinersen Versus 12/12mg Nusinersen
Description: as for outcome 39
Time Frame: Baseline, Day 302
Population: as for outcome 36
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Part B: Later-Onset SMA: 12/12 mg Nusinersen | Part B: Later-Onset SMA: 50/28 mg Nusinersen
Number analyzed (Participants) | 5 | 16
ratio | 0.28 [0.14 to 0.56] | 0.35 [0.24 to 0.51]

41. Secondary Outcome: Part B: Number of Participants With TEAEs and TESAEs
Description: AE was any unfavorable and unintended sign (including an abnormal assessment such as an abnormal laboratory value), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. An SAE was any untoward medical occurrence that at any dose resulted in death, in the view of the Investigator, placed the participant at immediate risk of death, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, resulted in a birth defect. AE was regarded as treatment-emergent if it was present prior to receiving the first dose of nusinersen in the current study and subsequently worsened in severity or was not present prior to receiving the first dose of nusinersen and subsequently appeared.
Time Frame: From the first dose of the study drug up to Day 399
Population: Safety set included all participants who received at least one dose of nusinersen.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Infantile-Onset SMA: 12/12 mg Nusinersen | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen | Part B: Later-Onset SMA: 12/12 mg Nusinersen | Part B: Later-Onset SMA: 50/28 mg Nusinersen
Number analyzed (Participants) | 25 | 50 | 8 | 16
Participants
  TEAEs | 22 | 45 | 7 | 14
  TESAEs | 18 | 30 | 4 | 2

42. Secondary Outcome: Part B: Number of Participants With Shifts From Baseline in Clinical Laboratory Parameters (Hematology Parameters)
Description: Hematology parameters included complete blood cell count, with diﬀerential and platelet count, and absolute neutrophil count. These parameters were flagged as low, normal, or high relative to parameter's normal range or as unknown if no result was available, by the Investigator. Here, shift to low indicates values that were normal, high or unknown at baseline and shifted to low values postbaseline. Shift to high indicates values that were normal, low or unknown at baseline and shifted to high values postbaseline. The categories with at least one participant with shift from baseline in these parameters are reported.
Time Frame: Baseline up to Day 302
Population: Safety set included all participants who received at least one dose of nusinersen. 'Number analysed (n)' signifies number of participants evaluable for analysis of the specified hematology parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Infantile-Onset SMA: 12/12 mg Nusinersen | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen | Part B: Later-Onset SMA: 12/12 mg Nusinersen | Part B: Later-Onset SMA: 50/28 mg Nusinersen
Number analyzed (Participants) | 25 | 50 | 8 | 16
Participants
  Basophils Shift to Low: number analyzed (Participants) | 22 | 46 | 8 | 16
  Basophils Shift to Low | 0 | 2 | 0 | 0
  Basophils Shift to High: number analyzed (Participants) | 12 | 24 | 5 | 13
  Basophils Shift to High | 7 | 17 | 4 | 8
  Basophils/Leukocytes Shift to High: number analyzed (Participants) | 11 | 21 | 4 | 9
  Basophils/Leukocytes Shift to High | 7 | 14 | 3 | 9
  Eosinophils Shift to Low: number analyzed (Participants) | 20 | 47 | 7 | 16
  Eosinophils Shift to Low | 0 | 7 | 1 | 0
  Eosinophils Shift to High: number analyzed (Participants) | 19 | 43 | 5 | 14
  Eosinophils Shift to High | 6 | 15 | 0 | 1
  Eosinophils/Leukocytes Shift to Low: number analyzed (Participants) | 21 | 47 | 8 | 16
  Eosinophils/Leukocytes Shift to Low | 0 | 4 | 0 | 0
  Eosinophils/Leukocytes Shift to High: number analyzed (Participants) | 15 | 28 | 5 | 12
  Eosinophils/Leukocytes Shift to High | 8 | 12 | 1 | 5
  Hematocrit Shift to Low: number analyzed (Participants) | 20 | 43 | 8 | 16
  Hematocrit Shift to Low | 6 | 12 | 0 | 2
  Hematocrit Shift to High: number analyzed (Participants) | 22 | 47 | 8 | 15
  Hematocrit Shift to High | 4 | 10 | 2 | 1
  Hemoglobin Shift to Low: number analyzed (Participants) | 22 | 45 | 7 | 14
  Hemoglobin Shift to Low | 11 | 18 | 0 | 2
  Hemoglobin Shift to High: number analyzed (Participants) | 23 | 46 | 8 | 16
  Hemoglobin Shift to High | 3 | 2 | 0 | 0
  Lymphocytes Shift to Low: number analyzed (Participants) | 22 | 47 | 8 | 16
  Lymphocytes Shift to Low | 3 | 6 | 1 | 1
  Lymphocytes Shift to High: number analyzed (Participants) | 19 | 41 | 7 | 14
  Lymphocytes Shift to High | 4 | 14 | 2 | 2
  Lymphocyte Atypical Shift to High: number analyzed (Participants) | 1 | 7 | 8 | 16
  Lymphocyte Atypical Shift to High | 0 | 5 | 0 | 0
  Lymphocyte Atypical/ Leukocyte Shift to High: number analyzed (Participants) | 1 | 7 | 8 | 16
  Lymphocyte Atypical/ Leukocyte Shift to High | 0 | 4 | 0 | 0
  Lymphocyte/Leukocyte Shift to Low: number analyzed (Participants) | 22 | 45 | 8 | 16
  Lymphocyte/Leukocyte Shift to Low | 4 | 5 | 1 | 2
  Lymphocyte/Leukocyte Shift to High: number analyzed (Participants) | 20 | 43 | 7 | 16
  Lymphocyte/Leukocyte Shift to High | 4 | 7 | 3 | 1
  Erythrocyte Mean Corpuscular Vol Shift to Low: number analyzed (Participants) | 5 | 10 | 8 | 16
  Erythrocyte Mean Corpuscular Vol Shift to Low | 2 | 2 | 0 | 0
  Erythrocyte Mean Corpuscular Vol Shift to High: number analyzed (Participants) | 4 | 8 | 8 | 16
  Erythrocyte Mean Corpuscular Vol Shift to High | 1 | 2 | 0 | 0
  Monocytes Shift to Low: number analyzed (Participants) | 22 | 46 | 7 | 15
  Monocytes Shift to Low | 5 | 12 | 1 | 6
  Monocytes Shift to High: number analyzed (Participants) | 20 | 42 | 8 | 16
  Monocytes Shift to High | 5 | 13 | 2 | 2
  Monocytes/Leukocytes Shift to Low: number analyzed (Participants) | 21 | 44 | 6 | 14
  Monocytes/Leukocytes Shift to Low | 7 | 20 | 1 | 9
  Monocytes/Leukocytes Shift to High: number analyzed (Participants) | 20 | 45 | 8 | 16
  Monocytes/Leukocytes Shift to High | 3 | 9 | 1 | 1
  Neutrophils Shift to Low: number analyzed (Participants) | 19 | 42 | 5 | 16
  Neutrophils Shift to Low | 5 | 9 | 1 | 2
  Neutrophils Shift to High: number analyzed (Participants) | 21 | 46 | 8 | 16
  Neutrophils Shift to High | 11 | 13 | 1 | 1
  Neutrophils/Leukocytes Shift to Low: number analyzed (Participants) | 19 | 39 | 7 | 16
  Neutrophils/Leukocytes Shift to Low | 4 | 13 | 4 | 0
  Neutrophils/Leukocytes Shift to High: number analyzed (Participants) | 21 | 45 | 7 | 16
  Neutrophils/Leukocytes Shift to High | 6 | 6 | 1 | 1
  Platelets Shift to Low: number analyzed (Participants) | 23 | 47 | 8 | 16
  Platelets Shift to Low | 1 | 2 | 0 | 1
  Platelets Shift to High: number analyzed (Participants) | 10 | 28 | 6 | 15
  Platelets Shift to High | 4 | 14 | 1 | 4
  Erythrocytes Shift to Low: number analyzed (Participants) | 23 | 46 | 6 | 15
  Erythrocytes Shift to Low | 4 | 10 | 0 | 0
  Erythrocytes Shift to High: number analyzed (Participants) | 22 | 47 | 8 | 13
  Erythrocytes Shift to High | 3 | 6 | 1 | 0
  Leukocytes Shift to Low: number analyzed (Participants) | 21 | 44 | 8 | 16
  Leukocytes Shift to Low | 4 | 13 | 2 | 0
  Leukocytes Shift to High: number analyzed (Participants) | 21 | 41 | 7 | 15
  Leukocytes Shift to High | 10 | 15 | 1 | 2

43. Secondary Outcome: Part B: Number of Participants With Shifts From Baseline in Clinical Laboratory Parameters (Blood Chemistry Parameters)
Description: Blood chemistry parameters included protein, albumin, creatinine, blood urea nitrogen, bilirubin (total and direct), alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase, gamma-glutamyl transferase, glucose, calcium, phosphorus, bicarbonate, chloride, sodium, potassium, cystatin C, and creatine kinase. Parameters were flagged as low, normal, or high relative to parameter's normal range or as unknown if no result was available, by the Investigator. Here, shift to low indicates values that were normal, high or unknown at baseline and shifted to low values postbaseline. Shift to high indicates values that were normal, low or unknown at baseline and shifted to high values postbaseline. Categories with at least one participant with shift from baseline in these parameters are reported.
Time Frame: Baseline up to Day 302
Population: Safety set included all participants who received at least one dose of nusinersen. 'Number analysed (n)' signifies number of participants evaluable for analysis of the specified parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Infantile-Onset SMA: 12/12 mg Nusinersen | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen | Part B: Later-Onset SMA: 12/12 mg Nusinersen | Part B: Later-Onset SMA: 50/28 mg Nusinersen
Number analyzed (Participants) | 25 | 50 | 8 | 16
Participants
  Albumin Shift to Low: number analyzed (Participants) | 20 | 46 | 8 | 15
  Albumin Shift to Low | 6 | 13 | 1 | 1
  Albumin Shift to High: number analyzed (Participants) | 23 | 50 | 8 | 16
  Albumin Shift to High | 1 | 2 | 0 | 0
  Alkaline Phosphatase Shift to Low: number analyzed (Participants) | 23 | 50 | 8 | 16
  Alkaline Phosphatase Shift to Low | 0 | 3 | 0 | 0
  Alkaline Phosphatase Shift to High: number analyzed (Participants) | 23 | 50 | 8 | 16
  Alkaline Phosphatase Shift to High | 3 | 3 | 0 | 0
  Alanine Aminotransferase Shift to Low: number analyzed (Participants) | 23 | 50 | 8 | 16
  Alanine Aminotransferase Shift to Low | 0 | 0 | 0 | 1
  Alanine Aminotransferase Shift to High: number analyzed (Participants) | 14 | 39 | 6 | 15
  Alanine Aminotransferase Shift to High | 4 | 14 | 0 | 3
  Aspartate Aminotransferase Shift to High: number analyzed (Participants) | 21 | 45 | 7 | 16
  Aspartate Aminotransferase Shift to High | 5 | 9 | 0 | 1
  Bicarbonate Shift to Low: number analyzed (Participants) | 5 | 14 | 3 | 4
  Bicarbonate Shift to Low | 4 | 12 | 3 | 4
  Bicarbonate Shift to High: number analyzed (Participants) | 22 | 49 | 8 | 16
  Bicarbonate Shift to High | 1 | 1 | 0 | 0
  Direct Bilirubin Shift to Low: number analyzed (Participants) | 22 | 45 | 8 | 16
  Direct Bilirubin Shift to Low | 1 | 0 | 0 | 0
  Bilirubin Shift to Low: number analyzed (Participants) | 21 | 49 | 8 | 16
  Bilirubin Shift to Low | 2 | 2 | 0 | 1
  Bilirubin Shift to High: number analyzed (Participants) | 20 | 45 | 8 | 16
  Bilirubin Shift to High | 1 | 1 | 0 | 0
  Indirect Bilirubin Shift to Low: number analyzed (Participants) | 22 | 46 | 2 | 4
  Indirect Bilirubin Shift to Low | 11 | 21 | 2 | 3
  Calcium Shift to Low: number analyzed (Participants) | 23 | 50 | 8 | 15
  Calcium Shift to Low | 1 | 4 | 2 | 1
  Calcium Shift to High: number analyzed (Participants) | 19 | 45 | 8 | 15
  Calcium Shift to High | 8 | 17 | 0 | 0
  Creatine Kinase Shift to High: number analyzed (Participants) | 14 | 27 | 6 | 10
  Creatine Kinase Shift to High | 6 | 12 | 3 | 3
  Chloride Shift to Low: number analyzed (Participants) | 23 | 50 | 8 | 16
  Chloride Shift to Low | 3 | 3 | 0 | 1
  Chloride Shift to High: number analyzed (Participants) | 23 | 48 | 7 | 16
  Chloride Shift to High | 3 | 6 | 1 | 1
  Creatinine Shift to Low | 2 | 5 | 0 | 1
  Creatinine Shift to High: number analyzed (Participants) | 23 | 50 | 8 | 16
  Creatinine Shift to High | 0 | 1 | 0 | 0
  Cystatin C Shift to Low: number analyzed (Participants) | 23 | 48 | 8 | 16
  Cystatin C Shift to Low | 2 | 0 | 1 | 1
  Cystatin C Shift to High: number analyzed (Participants) | 23 | 48 | 8 | 16
  Cystatin C Shift to High | 2 | 1 | 0 | 0
  Gamma Glutamyl Transferase Shift to Low: number analyzed (Participants) | 18 | 45 | 8 | 16
  Gamma Glutamyl Transferase Shift to Low | 7 | 11 | 0 | 1
  Gamma Glutamyl Transferase Shift to High: number analyzed (Participants) | 23 | 49 | 8 | 16
  Gamma Glutamyl Transferase Shift to High | 2 | 5 | 0 | 3
  Glucose Shift to Low: number analyzed (Participants) | 23 | 49 | 8 | 16
  Glucose Shift to Low | 0 | 2 | 0 | 1
  Glucose Shift to High: number analyzed (Participants) | 20 | 44 | 7 | 15
  Glucose Shift to High | 6 | 17 | 2 | 6
  Potassium Shift to Low: number analyzed (Participants) | 23 | 50 | 8 | 16
  Potassium Shift to Low | 1 | 2 | 0 | 1
  Potassium Shift to High: number analyzed (Participants) | 21 | 44 | 8 | 16
  Potassium Shift to High | 5 | 15 | 3 | 4
  Lactate Dehydrogenase Shift to High: number analyzed (Participants) | 25 | 1 | 8 | 16
  Lactate Dehydrogenase Shift to High | 0 | 1 | 0 | 0
  Magnesium Shift to High: number analyzed (Participants) | 3 | 50 | 8 | 16
  Magnesium Shift to High | 0 | 2 | 0 | 0
  Phosphate Shift to Low: number analyzed (Participants) | 23 | 50 | 8 | 16
  Phosphate Shift to Low | 3 | 2 | 0 | 0
  Phosphate Shift to High: number analyzed (Participants) | 18 | 42 | 4 | 13
  Phosphate Shift to High | 5 | 16 | 2 | 10
  Protein Shift to Low: number analyzed (Participants) | 21 | 48 | 7 | 15
  Protein Shift to Low | 7 | 9 | 1 | 2
  Protein Shift to High: number analyzed (Participants) | 23 | 47 | 8 | 16
  Protein Shift to High | 2 | 6 | 0 | 2
  Sodium Shift to Low: number analyzed (Participants) | 20 | 47 | 7 | 15
  Sodium Shift to Low | 3 | 15 | 2 | 3
  Sodium Shift to High: number analyzed (Participants) | 23 | 50 | 8 | 16
  Sodium Shift to High | 0 | 0 | 0 | 1
  Urea Nitrogen Shift to Low: number analyzed (Participants) | 23 | 44 | 8 | 16
  Urea Nitrogen Shift to Low | 1 | 3 | 2 | 1
  Urea Nitrogen Shift to High: number analyzed (Participants) | 23 | 50 | 8 | 15
  Urea Nitrogen Shift to High | 0 | 0 | 2 | 1

44. Secondary Outcome: Part B: Number of Participants With Shifts From Baseline in Urinalysis
Description: Urinalysis included assessments of urine total protein, specific gravity, pH, protein, glucose, ketones, bilirubin, blood, RBC , WBC, epithelial cells, bacteria, casts and crystals. These parameters were flagged as low, normal, or high relative to parameter's normal range or as unknown if no result was available, by the Investigator. Here, shift to low indicates values that were normal, high, positive, abnormal or unknown at baseline and shifted to low values postbaseline. Shift to high indicates values that were normal, negative, absent, low or unknown at baseline and shifted to high values postbaseline. The categories with at least one participant with shift from baseline in these parameters are reported.
Time Frame: Baseline up to Day 302
Population: as for outcome 43
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Infantile-Onset SMA: 12/12 mg Nusinersen | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen | Part B: Later-Onset SMA: 12/12 mg Nusinersen | Part B: Later-Onset SMA: 50/28 mg Nusinersen
Number analyzed (Participants) | 25 | 50 | 8 | 16
Participants
  Specific Gravity Shift to Low: number analyzed (Participants) | 20 | 47 | 8 | 16
  Specific Gravity Shift to Low | 2 | 2 | 1 | 1
  Specific Gravity Shift to High: number analyzed (Participants) | 22 | 50 | 7 | 15
  Specific Gravity Shift to High | 3 | 3 | 1 | 1
  pH Shift to Low: number analyzed (Participants) | 21 | 48 | 8 | 16
  pH Shift to Low | 2 | 1 | 0 | 1
  pH Shift to High: number analyzed (Participants) | 21 | 47 | 8 | 16
  pH Shift to High | 5 | 8 | 1 | 1
  Protein High/positive: number analyzed (Participants) | 18 | 45 | 5 | 13
  Protein High/positive | 12 | 27 | 3 | 9
  Glucose High/positive: number analyzed (Participants) | 21 | 46 | 8 | 16
  Glucose High/positive | 2 | 2 | 0 | 0
  Ketones High/positive: number analyzed (Participants) | 20 | 44 | 8 | 14
  Ketones High/positive | 5 | 16 | 4 | 4
  Occult Blood High/positive: number analyzed (Participants) | 16 | 43 | 7 | 14
  Occult Blood High/positive | 4 | 12 | 2 | 1
  RBC High/positive: number analyzed (Participants) | 13 | 26 | 7 | 12
  RBC High/positive | 0 | 3 | 0 | 0
  WBC High/positive: number analyzed (Participants) | 15 | 25 | 6 | 10
  WBC High/positive | 3 | 12 | 3 | 4
  Epithelial Cells High/positive: number analyzed (Participants) | 25 | 7 | 5 | 3
  Epithelial Cells High/positive | 0 | 6 | 5 | 2
  Bacteria High/positive: number analyzed (Participants) | 10 | 18 | 2 | 8
  Bacteria High/positive | 10 | 18 | 2 | 8
  Casts High/positive: number analyzed (Participants) | 3 | 3 | 8 | 16
  Casts High/positive | 0 | 1 | 0 | 0
  Crystals High/positive: number analyzed (Participants) | 5 | 4 | 8 | 16
  Crystals High/positive | 2 | 1 | 0 | 0

45. Secondary Outcome: Part B: Number of Participants With Shifts From Baseline in CSF Parameters
Description: as for outcome 6
Time Frame: Baseline up to Day 302
Population: Safety set included all participants who received at least one dose of nusinersen. 'Overall number of participants analyzed' signifies number of participants evaluable for this outcome measure. 'Number analysed (n)' signifies number of participants evaluable for analysis of the specified parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Infantile-Onset SMA: 12/12 mg Nusinersen | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen | Part B: Later-Onset SMA: 12/12 mg Nusinersen | Part B: Later-Onset SMA: 50/28 mg Nusinersen
Number analyzed (Participants) | 19 | 47 | 8 | 16
Participants
  Glucose Shift to Low: number analyzed (Participants) | 16 | 36 | 7 | 12
  Glucose Shift to Low | 4 | 3 | 1 | 0
  Glucose Shift to High: number analyzed (Participants) | 19 | 46 | 8 | 16
  Glucose Shift to High | 0 | 1 | 0 | 0
  Protein Shift to Low: number analyzed (Participants) | 18 | 45 | 5 | 11
  Protein Shift to Low | 2 | 6 | 0 | 4
  Protein Shift to High: number analyzed (Participants) | 12 | 25 | 8 | 15
  Protein Shift to High | 4 | 7 | 2 | 2
  Erythrocytes Shift to Low: number analyzed (Participants) | 18 | 47 | 8 | 15
  Erythrocytes Shift to Low | 1 | 0 | 0 | 0
  Erythrocytes Shift to High: number analyzed (Participants) | 14 | 37 | 5 | 11
  Erythrocytes Shift to High | 3 | 9 | 2 | 7
  Leukocytes Shift to Low: number analyzed (Participants) | 17 | 47 | 8 | 11
  Leukocytes Shift to Low | 1 | 2 | 0 | 1
  Leukocytes Shift to High: number analyzed (Participants) | 16 | 38 | 8 | 11
  Leukocytes Shift to High | 1 | 5 | 0 | 4

46. Secondary Outcome: Part B: Number of Participants With Shift From Baseline in ECGs
Description: as for outcome 7
Time Frame: Baseline up to Day 302
Population: Safety set included all participants who received at least one dose of nusinersen.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Infantile-Onset SMA: 12/12 mg Nusinersen | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen | Part B: Later-Onset SMA: 12/12 mg Nusinersen | Part B: Later-Onset SMA: 50/28 mg Nusinersen
Number analyzed (Participants) | 25 | 50 | 8 | 16
Participants
  Baseline: Normal; Postbaseline: Normal | 2 | 7 | 0 | 0
  Baseline: Normal ; Postbaseline: Abnormal, not AE | 9 | 10 | 2 | 4
  Baseline: Normal; Postbaseline: Abnormal, AE | 1 | 0 | 0 | 0
  Baseline: Abnormal, not AE; Postbaseline: Abnormal, not AE | 12 | 30 | 6 | 12
  Baseline: Abnormal, not AE; Postbaseline: Abnormal, AE | 1 | 2 | 0 | 0
  Baseline: Unknown; Postbaseline: Abnormal, not AE | 0 | 1 | 0 | 0

47. Secondary Outcome: Part B: Number of Participants With Abnormalities in Vital Sign Parameters
Description: Vital sign assessment included temperature, pulse rate systolic blood pressure, diastolic blood pressure, and respiratory rate. As pre-specified in protocol, the criteria for determining potentially clinically relevant abnormalities in vital signs included: temperature < 36.0 and > 38.0 degrees C, pulse rate < 60 and > 100 bpm, systolic blood pressure < 90, > 140 and > 160 mmHg, diastolic blood pressure < 50, > 90 and > 100 mmHg and respiratory rate < 12 and > 20 breaths per minute. The categories with at least one participant with clinically relevant vital sign abnormalities are reported.
Time Frame: Baseline up to Day 302
Population: as for outcome 43
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Infantile-Onset SMA: 12/12 mg Nusinersen | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen | Part B: Later-Onset SMA: 12/12 mg Nusinersen | Part B: Later-Onset SMA: 50/28 mg Nusinersen
Number analyzed (Participants) | 25 | 50 | 8 | 16
Participants
  Temperature <36.0 C | 6 | 23 | 3 | 7
  Temperature >38.0 C | 0 | 6 | 0 | 1
  Pulse Rate <60 bpm | 1 | 2 | 0 | 0
  Pulse Rate >100 bpm | 25 | 50 | 8 | 16
  Systolic Blood Pressure <90 mmHg: number analyzed (Participants) | 25 | 49 | 8 | 16
  Systolic Blood Pressure <90 mmHg | 24 | 47 | 7 | 10
  Systolic Blood Pressure >140 mmHg: number analyzed (Participants) | 25 | 49 | 8 | 16
  Systolic Blood Pressure >140 mmHg | 3 | 0 | 0 | 0
  Diastolic Blood Pressure <50 mmHg: number analyzed (Participants) | 25 | 49 | 8 | 16
  Diastolic Blood Pressure <50 mmHg | 22 | 44 | 4 | 10
  Diastolic Blood Pressure >90 mmHg: number analyzed (Participants) | 25 | 49 | 8 | 16
  Diastolic Blood Pressure >90 mmHg | 5 | 8 | 1 | 2
  Diastolic Blood Pressure >100 mmHg: number analyzed (Participants) | 25 | 49 | 8 | 16
  Diastolic Blood Pressure >100 mmHg | 0 | 0 | 0 | 1
  Respiratory Rate <12 breaths/min: number analyzed (Participants) | 25 | 49 | 8 | 16
  Respiratory Rate <12 breaths/min | 0 | 0 | 0 | 0
  Respiratory Rate >20 breaths/min | 25 | 50 | 8 | 16

48. Secondary Outcome: Part B: Change From Baseline in Growth Parameters (Body Height)
Description: Body height was measured for all participants (infantile-onset and later-onset SMA).
Time Frame: Baseline, Day 302
Population: Safety set included all participants who received at least one dose of nusinersen. 'Overall number of participants analyzed' signifies number of participants evaluable for this outcome measure at the specified time point.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Part B: Infantile-Onset SMA: 12/12 mg Nusinersen | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen | Part B: Later-Onset SMA: 12/12 mg Nusinersen | Part B: Later-Onset SMA: 50/28 mg Nusinersen
Number analyzed (Participants) | 1 | 4 | 1 | 8
cm | 8.0 (NA) — Since only one participant was evaluable SD was not estimable. | 10.25 (2.217) | 11.2 (NA) — Since only one participant was evaluable SD was not estimable. | 6.9 (3.65)

49. Secondary Outcome: Part B Infantile-onset SMA: Change From Baseline in Growth Parameters (Head Circumference)
Description: Head circumference was measured in participants with infantile-onset SMA.
Time Frame: Baseline, Day 302
Population: as for outcome 48
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Part B: Infantile-Onset SMA: 12/12 mg Nusinersen | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen
Number analyzed (Participants) | 13 | 35
cm | 4.52 (1.703) | 5.50 (2.766)

50. Secondary Outcome: Part B Infantile-onset SMA: Change From Baseline in Growth Parameters (Chest Circumference)
Description: Chest circumference was measured in participants with infantile-onset SMA.
Time Frame: Baseline, Day 302
Population: as for outcome 48
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Part B: Infantile-Onset SMA: 12/12 mg Nusinersen | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen
Number analyzed (Participants) | 13 | 35
cm | 5.67 (4.868) | 6.64 (6.362)

51. Secondary Outcome: Part B Infantile-onset SMA: Change From Baseline in Growth Parameters (Arm Circumference)
Description: Arm circumference was measured in participants with infantile-onset SMA.
Time Frame: Baseline, Day 302
Population: as for outcome 48
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Part B: Infantile-Onset SMA: 12/12 mg Nusinersen | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen
Number analyzed (Participants) | 13 | 35
cm | 0.45 (2.141) | 1.16 (2.144)

52. Secondary Outcome: Part B: Change From Baseline in Growth Parameters (Ulnar Length)
Description: Ulnar length was measured in participants with later-onset SMA.
Time Frame: Baseline, Day 302
Population: as for outcome 48
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Part B: Later-Onset SMA: 12/12 mg Nusinersen | Part B: Later-Onset SMA: 50/28 mg Nusinersen
Number analyzed (Participants) | 5 | 16
cm | 2.8 (4.16) | 1.2 (1.39)

53. Secondary Outcome: Part B: Change From Baseline in Growth Parameters (Weight for Age Percentile)
Description: WHO child growth standards (2006) was used to calculate the weight for age percentile in the infantile-onset participants. The 2000 CDC Growth Charts was used to calculate the weight for age percentile for later-onset participants. Negative change from baseline indicates reduction in weight for age percentile
Time Frame: Baseline, Day 302
Population: as for outcome 48
Measure: Mean (Standard Deviation); unit: percentile
Arm/Group | Part B: Infantile-Onset SMA: 12/12 mg Nusinersen | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen | Part B: Later-Onset SMA: 12/12 mg Nusinersen | Part B: Later-Onset SMA: 50/28 mg Nusinersen
Number analyzed (Participants) | 13 | 35 | 7 | 16
percentile | -6.70 (23.133) | -3.60 (35.202) | 9.1 (20.23) | -0.3 (6.96)

54. Secondary Outcome: Part B: Change From Baseline in Growth Parameters (Weight for Length Percentile)
Description: As pre-specified in the protocol, weight for length percentile was assessed only for the participants with infantile-onset SMA. Negative change from baseline indicates reduction in weight for length percentile.
Time Frame: Baseline, Day 302
Population: as for outcome 48
Measure: Mean (Standard Deviation); unit: percentile
Arm/Group | Part B: Infantile-Onset SMA: 12/12 mg Nusinersen | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen
Number analyzed (Participants) | 12 | 30
percentile | -4.23 (35.817) | 6.05 (40.119)

55. Secondary Outcome: Part B: Change From Baseline in Growth Parameters (Head-to-Chest Circumference Ratio)
Description: As pre-specified in the protocol, head to chest circumference ratio was assessed only for the participants with infantile-onset SMA. Negative change from baseline indicates reduction in head-to-chest circumference ratio.
Time Frame: Baseline, Day 302
Population: as for outcome 48
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Part B: Infantile-Onset SMA: 12/12 mg Nusinersen | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen
Number analyzed (Participants) | 13 | 35
ratio | -0.03 (0.085) | -0.05 (0.269)

56. Secondary Outcome: Part B: Number of Participants With Shifts From Baseline in Coagulation Parameters (aPTT)
Description: aPTT was evaluated to assess safety. "Shift to low" measured change in normal, high and unknown values of aPTT at baseline to low values postbaseline. "Shift to high" measured change in normal, low and unknown values of aPTT at baseline to high values postbaseline.
Time Frame: Baseline up to Day 279
Population: Safety set included all participants who received at least one dose of nusinersen. 'Number analysed (n)' signifies number of participants evaluable for the specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Infantile-Onset SMA: 12/12 mg Nusinersen | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen | Part B: Later-Onset SMA: 12/12 mg Nusinersen | Part B: Later-Onset SMA: 50/28 mg Nusinersen
Number analyzed (Participants) | 25 | 50 | 8 | 16
Participants
  Shift to Low: number analyzed (Participants) | 22 | 48 | 7 | 16
  Shift to Low | 4 | 14 | 2 | 2
  Shift to High: number analyzed (Participants) | 17 | 40 | 8 | 15
  Shift to High | 6 | 7 | 1 | 1

57. Secondary Outcome: Part B: Number of Participants With Shifts From Baseline in Coagulation Parameters (PT)
Description: as for outcome 18
Time Frame: Baseline up to Day 279
Population: as for outcome 56
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Infantile-Onset SMA: 12/12 mg Nusinersen | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen | Part B: Later-Onset SMA: 12/12 mg Nusinersen | Part B: Later-Onset SMA: 50/28 mg Nusinersen
Number analyzed (Participants) | 25 | 50 | 8 | 16
Participants
  Shift to Low: number analyzed (Participants) | 22 | 48 | 8 | 15
  Shift to Low | 3 | 6 | 1 | 1
  Shift to High: number analyzed (Participants) | 20 | 45 | 8 | 14
  Shift to High | 2 | 6 | 0 | 1

58. Secondary Outcome: Part B: Number of Participants With Shifts From Baseline in Coagulation Parameters (INR)
Description: INR was evaluated to assess safety. "Shift to low" measured change in normal, high and unknown values of INR at baseline to low values postbaseline. "Shift to high" measured change in normal, low and unknown values of INR at baseline to high values postbaseline.
Time Frame: Baseline up to Day 279
Population: as for outcome 56
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Infantile-Onset SMA: 12/12 mg Nusinersen | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen | Part B: Later-Onset SMA: 12/12 mg Nusinersen | Part B: Later-Onset SMA: 50/28 mg Nusinersen
Number analyzed (Participants) | 25 | 50 | 8 | 16
Participants
  Shift to Low: number analyzed (Participants) | 22 | 49 | 8 | 16
  Shift to Low | 1 | 5 | 0 | 0
  Shift to High: number analyzed (Participants) | 21 | 44 | 8 | 16
  Shift to High | 2 | 6 | 1 | 0

59. Secondary Outcome: Part B: Change From Baseline in Urine Total Protein
Time Frame: Baseline, Day 302
Population: Safety set included all participants who received at least one dose of nusinersen. 'Overall number of participants analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | Part B: Infantile-Onset SMA: 12/12 mg Nusinersen | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen | Part B: Later-Onset SMA: 12/12 mg Nusinersen | Part B: Later-Onset SMA: 50/28 mg Nusinersen
Number analyzed (Participants) | 7 | 18 | 3 | 11
grams per liter (g/L) | -0.130 (0.4126) | -3.274 (14.1387) | -0.213 (0.2873) | 0.004 (0.0608)

60. Secondary Outcome: Part B: Number of Participants With Neurological Examination Abnormalities Reported as AEs
Description: Participants with abnormalities in neurological examinations recorded as AEs were reported.
Time Frame: Baseline up to Day 302
Population: Safety set included all participants who received at least one dose of nusinersen.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Infantile-Onset SMA: 12/12 mg Nusinersen | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen | Part B: Later-Onset SMA: 12/12 mg Nusinersen | Part B: Later-Onset SMA: 50/28 mg Nusinersen
Number analyzed (Participants) | 25 | 50 | 8 | 16
Participants
  Muscular Weakness | 0 | 1 | 0 | 0
  Bulbar Palsy | 1 | 0 | 0 | 0
  Tremor | 0 | 0 | 0 | 1

61. Secondary Outcome: Part B: Percentage of Participants With a Postbaseline Platelet Count Below the Lower Limit of Normal on at Least 2 Consecutive Measurements
Time Frame: Baseline up to Day 302
Population: Safety set included all participants who received at least one dose of nusinersen.
Measure: Number; unit: percentage of participants
Arm/Group | Part B: Infantile-Onset SMA: 12/12 mg Nusinersen | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen | Part B: Later-Onset SMA: 12/12 mg Nusinersen | Part B: Later-Onset SMA: 50/28 mg Nusinersen
Number analyzed (Participants) | 25 | 50 | 8 | 16
percentage of participants | 4 | 0 | 0 | 0

62. Secondary Outcome: Part B: Percentage of Participants With a Postbaseline QTcF of > 500 Msec and an Increase From Baseline to Any Postbaseline Timepoint in QTcF of > 60 Msec
Time Frame: Baseline up to Day 302
Population: as for outcome 59
Measure: Number; unit: percentage of participants
Arm/Group | Part B: Infantile-Onset SMA: 12/12 mg Nusinersen | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen | Part B: Later-Onset SMA: 12/12 mg Nusinersen | Part B: Later-Onset SMA: 50/28 mg Nusinersen
Number analyzed (Participants) | 25 | 49 | 8 | 16
percentage of participants | 8 | 0 | 0 | 0

63. Secondary Outcome: Parts A, B and C: Number of Participants With Hospitalizations
Time Frame: Parts A, B, and C: Baseline up to Day 302
Population: Parts A, B and C: ITT set included all participants who received at least one dose of nusinersen in the current study.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Nusinersen 28/28 mg | Part B: Infantile-Onset SMA: 12/12 mg Nusinersen | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen | Part B: Later-Onset SMA: 12/12 mg Nusinersen | Part B: Later-Onset SMA: 50/28 mg Nusinersen | Part C: Nusinersen 50/28 mg
Number analyzed (Participants) | 6 | 25 | 50 | 8 | 16 | 40
Participants | 1 | 19 | 26 | 3 | 6 | 12

64. Secondary Outcome: Parts A, B and C: Percentage of Time of Hospitalization
Time Frame: Parts A, B, and C: Baseline up to Day 302
Population: Parts A, B and C: ITT set included all participants who received at least one dose of nusinersen in the current study.
Measure: Median (Full Range); unit: percentage of days
Arm/Group | Part A: Nusinersen 28/28 mg | Part B: Infantile-Onset SMA: 12/12 mg Nusinersen | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen | Part B: Later-Onset SMA: 12/12 mg Nusinersen | Part B: Later-Onset SMA: 50/28 mg Nusinersen | Part C: 50/28 mg Nusinersen
Number analyzed (Participants) | 6 | 25 | 50 | 8 | 16 | 40
percentage of days | 0 [0 to 2] | 6.4 [0 to 100] | 1.9 [0 to 100] | 0.0 [0 to 8] | 0.0 [0 to 11] | 1.34 [0.3 to 10.4]

65. Secondary Outcome: Parts A, B and C: Number of Participants With Clinical Global Impression of Change (CGIC)
Description: The CGIC scale was a 7 point scale that required the clinician to assess how much the participant's illness had changed relative to a baseline state at the beginning of the intervention, where 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, 7=very much worse. Higher rating indicates worsening of the condition. A separate CGIC assessment was performed by the Investigator (I) and caregiver (C). The categories with at least one participant having a CGIC score was reported.
Time Frame: Parts A, B, and C: Day 302
Population: ITT set included all participants who received at least one dose of nusinersen in the current study. 'Overall number of participants analyzed' signifies number of participants evaluable for this outcome measure. 'Number analyzed' indicates the number of participants evaluable for the specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Nusinersen 28/28 mg | Part B: Infantile-Onset SMA: 12/12 mg Nusinersen | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen | Part B: Later-Onset SMA: 12/12 mg Nusinersen | Part B: Later-Onset SMA: 50/28 mg Nusinersen | Part C: 50/28 mg Nusinersen
Number analyzed (Participants) | 6 | 13 | 35 | 7 | 16 | 40
Participants
  CGIC-I: Very Much Improved | 0 | 0 | 8 | 0 | 1 | 0
  CGIC-I: Much Improved | 1 | 10 | 20 | 3 | 5 | 5
  CGIC-I: Minimally Improved | 5 | 3 | 7 | 4 | 9 | 19
  CGIC-I: No Change | 0 | 0 | 0 | 0 | 1 | 14
  CGIC-I: Minimally Worse | 0 | 0 | 0 | 0 | 0 | 2
  CGIC-C: number analyzed (Participants) | 6 | 13 | 35 | 7 | 16 | 24
  CGIC-C: Very Much Improved | 1 | 3 | 18 | 1 | 0 | 2
  CGIC-C: Much Improved | 2 | 7 | 13 | 2 | 8 | 6
  CGIC-C: Minimally Improved | 2 | 3 | 3 | 4 | 7 | 9
  CGIC-C: No Change | 0 | 0 | 1 | 0 | 1 | 5
  CGIC-C: Minimally Worse | 1 | 0 | 0 | 0 | 0 | 2

66. Secondary Outcome: Parts A, B and C: Number of Serious Respiratory Events
Time Frame: Parts A, B, and C: Baseline up to Day 399
Population: ITT set included all participants who received at least one dose of nusinersen in the current study.
Measure: Number; unit: number of events
Arm/Group | Part A: Nusinersen 28/28 mg | Part B: Infantile-Onset SMA: 12/12 mg Nusinersen | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen | Part B: Later-Onset SMA: 12/12 mg Nusinersen | Part B: Later-Onset SMA: 50/28 mg Nusinersen | Part C: 50/28 mg Nusinersen
Number analyzed (Participants) | 6 | 25 | 50 | 8 | 16 | 40
number of events | 0 | 34 | 60 | 6 | 2 | 0

67. Secondary Outcome: Part B Infantile-onset SMA: Percentage of Time on Ventilation
Time Frame: Baseline up to Day 302
Population: ITT set included all participants who were randomized and received at least one dose of nusinersen.
Measure: Median (Full Range); unit: percentage of hours
Arm/Group | Part B: Infantile-Onset SMA: 12/12 mg Nusinersen | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen
Number analyzed (Participants) | 25 | 50
percentage of hours | 5.6 [0 to 100] | 7.5 [0 to 100]

68. Secondary Outcome: Parts A, B and C: Number of Participants With Ventilator Use
Time Frame: Parts A, B, and C: Screening up to Day 302
Population: ITT set included all participants who received at least one dose of nusinersen in the current study.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Nusinersen 28/28 mg | Part B: Infantile-Onset SMA: 12/12 mg Nusinersen | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen | Part B: Later-Onset SMA: 12/12 mg Nusinersen | Part B: Later-Onset SMA: 50/28 mg Nusinersen | Part C: 50/28 mg Nusinersen
Number analyzed (Participants) | 6 | 25 | 50 | 8 | 16 | 40
Participants | 0 | 9 | 22 | 4 | 5 | 8

69. Secondary Outcome: Part A: Change From Baseline in the Parent Assessment of Swallowing Ability (PASA) Scale
Description: PASA was assessed using a questionnaire. Caregivers were asked a series of questions regarding the mealtime behavior of the participant. The PASA questionnaire was developed to assess the signs and symptoms of dysphagia. It included 33 items across 4 domains: general feeding, drinking liquids, eating solid foods, & assessment of swallowing concerns. Items in domains general feeding, drinking liquids, & eating solid foods are assessed with 5 levels of response scored as 4-Never, 3-Rarely, 2-Sometimes, 1-Often, & 0-Always. Domain for assessing swallowing concerns has 4 levels of responses scored as: 3-Strongly Disagree, 2-Disagree, 1-Agree, 0-Strongly Agree. Higher score= improvement. A negative change from baseline=decrease in swallowing ability. From domains 'drinking liquids' and 'eating solid foods', 2 items (attempted to drink liquids and eat solid foods) were assessed as "Yes"/"No", which are reported in another outcome measure.
Time Frame: Baseline, Day 302
Population: ITT set included all participants who received at least one dose of nusinersen. 'Number analysed (n)' signifies the number of participants evaluable for the specified parameter.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Part A: Nusinersen 28/28 mg
Number analyzed (Participants) | 6
score on scale
  Had Difficulty Feeding Themselves | 0.2 (0.41)
  Had to Suction Excess Saliva/Drool | 0.0 (0.00)
  Not Able Eat as Much as Would Like | 0.2 (0.41)
  Not Able Eat Food Variety Would Like | -0.2 (0.41)
  Been Tube-Fed | 0.0 (0.00)
  Refused Liquid Foods: number analyzed (Participants) | 4
  Refused Liquid Foods | 0.0 (0.00)
  Difficulty Drinking Thin Liquids: number analyzed (Participants) | 4
  Difficulty Drinking Thin Liquids | 0.0 (0.00)
  Difficulty Drinking Thick Liquids: number analyzed (Participants) | 4
  Difficulty Drinking Thick Liquids | 0.0 (0.00)
  Cough/Clear Throat Swallow Liquid Food: number analyzed (Participants) | 4
  Cough/Clear Throat Swallow Liquid Food | 0.0 (0.00)
  Gagged or Choked on Liquid Food: number analyzed (Participants) | 4
  Gagged or Choked on Liquid Food | 0.0 (0.00)
  Retching/Vomiting Drinking Liquids: number analyzed (Participants) | 4
  Retching/Vomiting Drinking Liquids | 0.0 (0.00)
  Taken > 30 Minutes Drink Liquids: number analyzed (Participants) | 4
  Taken > 30 Minutes Drink Liquids | 0.0 (0.00)
  Refused Solid Foods | 0.2 (0.41)
  Difficulty Swallowing Soft Foods | 0.0 (0.00)
  Difficulty Swallowing Solid Foods | -0.2 (0.41)
  Had Difficulty Swallowing Pills | 0.2 (0.98)
  Cough/Clear Throat Eat/Swallow Solid Food | 0.2 (0.41)
  Had Food Stuck in Throat/Chest | 0.0 (0.00)
  Gagged/Choked on Their Solid Food | 0.2 (0.41)
  Retching/Vomiting Eating Solids | 0.2 (0.41)
  Required Food to Be Cut Up | 0.7 (1.21)
  Experienced/Shown Pain When Eating | 0.0 (0.00)
  Has Taken > 30 Minutes Eat Solids | 0.3 (0.52)
  Concern Child's Swallowing Ability | 0.8 (1.72)
  Concerned About Child's Weight | 1.2 (1.60)
  Concern Variety Foods Child Eats | 0.7 (1.51)
  Concern Child Not Able Eat as Much | 1.3 (1.51)
  Concern Child Unable Eat Variety | 1.3 (1.37)
  Concern Not Get Goodness From Diet | 1.8 (1.17)
  Concerned Child Aspirating Food | 1.0 (1.55)
  Concern Child Choking When Eating | 1.2 (1.60)

70. Secondary Outcome: Part A: Number of Participants With Shift From Baseline in PASA Scale Items - Attempted to Drink Liquids and Attempted to Eat Solid Foods
Description: PASA was assessed using a questionnaire. Caregivers were asked a series of questions regarding the mealtime behavior of the participant. The PASA questionnaire was developed to assess the signs and symptoms of dysphagia. It included 33 items across 4 domains that cover general feeding, drinking liquids, eating solid foods, and assessment of swallowing concerns. The 2 items of domains drinking liquids (attempted to drink liquids), eating solid foods (attempted to eat solid foods) were assessed as "Yes"/"No". Data for the 2 items were summarized in terms of the shift from baseline.
Time Frame: Baseline, Day 302
Population: ITT set included all participants who received at least one dose of nusinersen.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Nusinersen 28/28 mg
Number analyzed (Participants) | 6
Participants
  Attempted to Drink Liquid Foods: Baseline: No, Post-baseline: Yes | 0 [lower limit 0.00]
  Attempted to Drink Liquid Foods: Baseline: No, Post-baseline: No | 2 [lower limit 0.00]
  Attempted to Drink Liquid Foods: Baseline: Yes, Post-baseline: Yes | 4 [lower limit 0.00]
  Attempted to Drink Liquid Foods: Baseline: Yes, Post-baseline: No | 0 [lower limit 0.00]
  Attempted to Eat Solid Foods: Baseline: No, Post-baseline: Yes | 0 [lower limit 0.00]
  Attempted to Eat Solid Foods: Baseline: No, Post-baseline: No | 0 [lower limit 0.00]
  Attempted to Eat Solid Foods: Baseline: Yes, Post-baseline: Yes | 6 [lower limit 0.00]
  Attempted to Eat Solid Foods: Baseline: Yes, Post-baseline: No | 0 [lower limit 0.00]

71. Secondary Outcome: Part B: Change From Baseline in the PASA Scale
Description: PASA was assessed using a questionnaire. Caregivers were asked a series of questions regarding the mealtime behavior of the participant. The PASA questionnaire was developed to assess the signs and symptoms of dysphagia. It included 33 items across 4 domains that cover general feeding, drinking liquids, eating solid foods, and assessment of swallowing concerns. Items in domains of general feeding, drinking liquids, & eating solid foods are assessed with 5 levels of response scored as 4-Never, 3-Rarely, 2-Sometimes, 1-Often, & 0-Always. Domain for assessing swallowing concerns has 4 levels of responses scored as: 3-Strongly Disagree, 2-Disagree, 1-Agree, 0-Strongly Agree. Higher score= improvement. A negative change from baseline=decrease in swallowing ability. As planned, for part B of the study, the PASA scale was assessed for the domain general feeding only.
Time Frame: Baseline, Day 302
Population: ITT set included all participants who were randomized and received at least one dose of nusinersen. 'Overall number of participants analyzed' signifies number of participants evaluable for this outcome measure. 'Number analysed (n)', signifies the number of participants evaluable for the specified parameter.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Part B: Infantile-Onset SMA: 12/12 mg Nusinersen | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen | Part B: Later-Onset SMA: 12/12 mg Nusinersen | Part B: Later-Onset SMA: 50/28 mg Nusinersen
Number analyzed (Participants) | 9 | 32 | 7 | 14
score on scale
  Had Difficulty Feeding Themselves: number analyzed (Participants) | 7 | 29 | 7 | 14
  Had Difficulty Feeding Themselves | -1.6 (1.81) | -0.6 (1.55) | -0.4 (0.53) | 0.3 (0.73)
  Had To Suction Excess Saliva or Drool: number analyzed (Participants) | 7 | 31 | 7 | 14
  Had To Suction Excess Saliva or Drool | -1.7 (1.38) | -0.2 (1.58) | 0.1 (0.38) | 0.1 (0.36)
  Not Able To Eat As Much As Would Like: number analyzed (Participants) | 7 | 31 | 7 | 14
  Not Able To Eat As Much As Would Like | -1.6 (1.72) | -0.2 (1.45) | 0.3 (0.95) | 0.0 (0.39)
  Not Able To Eat Food Variety They Like: number analyzed (Participants) | 7 | 29 | 7 | 14
  Not Able To Eat Food Variety They Like | -1.6 (1.72) | -1.0 (1.18) | 0.1 (0.69) | -0.4 (0.93)
  Been Tube-Fed | -1.8 (2.11) | -0.9 (1.76) | 0.0 (0.00) | 0.0 (0.00)

72. Secondary Outcome: Part B: Infantile SMA-onset: Change From (Ratio to) Baseline in CSF Concentration of NF-L
Description: as for outcome 39
Time Frame: Baseline, Day 279
Population: ITT set included all participants who were randomized and received at least one dose of nusinersen.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Part B: Infantile-Onset SMA: 12/12 mg Nusinersen | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen
Number analyzed (Participants) | 25 | 50
ratio | 0.06 [0.05 to 0.08] | 0.05 [0.04 to 0.06]
Statistical Analysis 1: Comparison: Part B: Infantile-Onset SMA: 12/12 mg Nusinersen vs Part B: Infantile-Onset SMA: 50/28 mg Nusinersen; Test type: Superiority; p = 0.3785, ANCOVA — ANCOVA model was used with treatment as a fixed effect and adjusted for each participant disease duration at screening, baseline log CSF NF-L and baseline CHOP INTEND total score; LS geometric mean ratio = 0.86, 95% CI 2-sided [0.62 to 1.2]

73. Secondary Outcome: Parts A and C: Change From Baseline in HFMSE Total Score
Description: HFMSE scale was a tool used to assess motor function in children with SMA. The original 20 item Hammersmith Functional Motor Scale was expanded to include 13 additional adapted items from the Gross Motor Function Measure to improve sensitivity for the higher functioning ambulant population. Each item is scored 0 (unable), 1 (performs with modification or adaptation) or 2 (able) and the total score was calculated by summing the 33 items and ranged from 0 to 66 with higher scores indicating greater motor function. Negative change from baseline indicates decrease in motor function.
Time Frame: Parts A and C: Baseline, Day 302
Population: ITT set included all participants who received at least one dose of nusinersen in the current study. 'Overall number of participants analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Part A: Nusinersen 28/28 mg | Part C: 50/28 mg Nusinersen
Number analyzed (Participants) | 6 | 38
score on scale | -0.8 (3.76) | 1.8 (3.99)

74. Secondary Outcome: Parts A and C: Change From Baseline in RULM Total Score
Description: as for outcome 35
Time Frame: Parts A and C: Baseline, Day 302
Population: as for outcome 73
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Part A: Nusinersen 28/28 mg | Part C: 50/28 mg Nusinersen
Number analyzed (Participants) | 6 | 37
score on scale | 1.5 (1.52) | 1.2 (2.14)

75. Secondary Outcome: Parts A and C: Number of Participants With WHO Motor Milestones Status
Description: The WHO motor milestones were a set of six milestones in motor development: sitting without support, standing with assistance, hands and knees crawling, walking with assistance, standing alone and walking alone. The examiner recorded an overall rating of the participant's emotional state and then for each milestone one of the following four classifications: no (inability) - child tried but failed to perform the milestone, no (refusal) - child refused to perform despite being calm and alert, yes - child was able to perform the milestone, unable to test - could not be tested because of irritability, drowsiness or sickness.
Time Frame: Parts A and C: Baseline up to Day 302
Population: as for outcome 73
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Nusinersen 28/28 mg | Part C: 50/28 mg Nusinersen
Number analyzed (Participants) | 6 | 37
Participants
  Gain of one or More Motor Milestones | 0 | 3
  No Change | 6 | 32
  Loss of one or More Motor Milestones | 0 | 2

76. Secondary Outcome: Parts A and C: Change From Baseline in ACEND Total Score
Description: as for outcome 37
Time Frame: Parts A and C: Baseline, Day 302
Population: as for outcome 73
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Part A: Nusinersen 28/28 mg | Part C: 50/28 mg Nusinersen
Number analyzed (Participants) | 6 | 17
score on scale
  Feeding/Grooming/Dressing Total Score | 0.6 (2.51) | 0.8 (7.50)
  Sitting/Play Total Score | 0.0 (11.03) | -2.8 (14.48)
  Transfers Total Score | -8.0 (12.39) | -2.0 (15.34)
  Mobility Total Score | 7.1 (13.85) | -0.8 (15.01)
  Time Total Score | 6.3 (14.25) | 0.4 (10.47)
  Emotion Total Score | 11.1 (7.66) | -2.4 (9.44)
  Finance Total Score | 15.8 (14.29) | -2.4 (12.00)

77. Secondary Outcome: Parts A and C: Change From Baseline in PedsQL™ Total Score
Description: as for outcome 38
Time Frame: Parts A and C: Baseline, Day 302
Population: ITT set included all participants who received at least one dose of nusinersen in the current study. 'Overall number of participants analyzed' signifies number of participants evaluable for this outcome measure. 'Number analysed (n)' signifies number of participants evaluable for the specified total score.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Part A: Nusinersen 28/28 mg | Part C: 50/28 mg Nusinersen
Number analyzed (Participants) | 6 | 14
score on scale
  PQLI-Total Score-Participant: number analyzed (Participants) | 5 | 12
  PQLI-Total Score-Participant | 6.1 (18.228) | 1.1 (9.74)
  PQLI-Total Score-Parent: number analyzed (Participants) | 5 | 14
  PQLI-Total Score-Parent | 3.3 (12.51) | 0.7 (8.15)
  PQLN-Total Score-Participant: number analyzed (Participants) | 5 | 12
  PQLN-Total Score-Participant | 9.9 (6.94) | 6.7 (13.11)
  PQLN-Total Score-Parent: number analyzed (Participants) | 6 | 13
  PQLN-Total Score-Parent | 4.7 (5.72) | 0.1 (9.65)

78. Secondary Outcome: Part C: Change From Baseline in CHOP-INTEND Total Score
Description: The CHOP-INTEND test was designed to evaluate the motor skills of infants with significant motor weakness. It included 16 items (capturing neck, trunk, and proximal and distal limb strength), nine of which were scored 0, 1, 2, 3, or 4, five were scored as 0, 2, or 4, one was scored as 0, 1, 2, or 4, and one as 0, 2, 3, or 4 with higher scores indicating greater muscle strength and function. Total score was calculated as the sum of scores for each item. Total score ranged from 0 (worst possible score) and 64 (best possible score).
Time Frame: Baseline, Day 302
Population: ITT set included all participants who received at least one dose of nusinersen in the current study. It was planned to be assessed in infantile-onset SMA participants. 'Overall number of participants analyzed' signifies number of participants with data available for outcome measure analysis.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Part C: 50/28 mg Nusinersen
Number analyzed (Participants) | 1
score on scale | 0.0 (NA) — Since only one participant was evaluable SD was not estimable.

79. Secondary Outcome: Part C: Change From Baseline in HINE Section 2 Motor Milestones Total Score
Description: Section 2 of the HINE was used to assess motor milestones of the infantile-onset SMA participants. It's composed of 8 motor milestone categories: voluntary grasp, ability to kick in supine position, head control, rolling, sitting, crawling, standing, and walking. Within each of these categories, participants can progress from complete absence of a motor ability (the lowest level in each category) through multiple milestones (2 to 4 levels in each category) to the highest level within the category. The 8 categories of HINE Section 2 can be summed to give a total score that ranges from 0 to 26.
Time Frame: Baseline, Day 302
Population: ITT set included all participants who received at least one dose of nusinersen in the current study. It was planned to be assessed in infantile-onset SMA participants. 'Overall number of participants analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Part C: 50/28 mg Nusinersen
Number analyzed (Participants) | 1
score on scale | 2.0 (NA) — Since only one participant was evaluable SD was not estimable.

ADVERSE EVENTS:
Time Frame: Part A: From first dose of the study up to Day 389 Part B: From first dose of the study up to Day 399 Part C: From first dose of the study up to Day 361
Description: Safety set included all participants who received at least one dose of nusinersen in this study. MedDRA version 24.0 was applied for Part A, MedDRA version 26.1 was applied for Part B, and MedDRA version 26.0 was applied for Part C.
Arm/Group | Part A: 28/28 mg Nusinersen | Part B: Infantile-Onset SMA: 12/12 mg Nusinersen | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen | Part B: Later-Onset SMA: 12/12 mg Nusinersen | Part B: Later-Onset SMA: 50/28 mg Nusinersen | Part C: 50/28 mg Nusinersen
All-Cause Mortality (participants affected / at risk) | 0/6 | 6/25 | 10/50 | 0/8 | 0/16 | 0/40
Serious Adverse Events (participants affected / at risk) | 1/6 | 18/25 | 30/50 | 4/8 | 2/16 | 6/40
Other Adverse Events (participants affected / at risk) | 4/6 | 19/25 | 37/50 | 7/8 | 14/16 | 36/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: 28/28 mg Nusinersen (N=6) | Part B: Infantile-Onset SMA: 12/12 mg Nusinersen (N=25) | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen (N=50) | Part B: Later-Onset SMA: 12/12 mg Nusinersen (N=8) | Part B: Later-Onset SMA: 50/28 mg Nusinersen (N=16) | Part C: 50/28 mg Nusinersen (N=40)
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 2
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 2
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Organ failure (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sudden infant death syndrome (General disorders) | 0 | 1 | 2 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 2 | 3 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 2 | 0 | 0 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Adenoviral upper respiratory infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 1 | 3 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 0 | 0 | 3 | 0 | 1 | 0
Enterovirus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis adenovirus (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis Escherichia coli (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Human coronavirus OC43 infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Lower respiratory tract infection viral (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Measles (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Norovirus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 5 | 7 | 0 | 0 | 0
Pneumonia acinetobacter (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia aspiration (Infections and infestations) | 0 | 1 | 7 | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Pneumonia influenzal (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Pneumonia mycoplasmal (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Pneumonia pseudomonal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 0
Pneumonia viral (Infections and infestations) | 0 | 1 | 2 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0
Rhinovirus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Stoma site infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Gastroenteritis rotavirus (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Acquired macrocephaly (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Brain stem infarction (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypoglycaemic seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 0 | 0
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 8 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: 28/28 mg Nusinersen (N=6) | Part B: Infantile-Onset SMA: 12/12 mg Nusinersen (N=25) | Part B: Infantile-Onset SMA: 50/28 mg Nusinersen (N=50) | Part B: Later-Onset SMA: 12/12 mg Nusinersen (N=8) | Part B: Later-Onset SMA: 50/28 mg Nusinersen (N=16) | Part C: 50/28 mg Nusinersen (N=40)
Headache (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 5
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bulbar palsy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Febrile convulsion (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2 | 4 | 1 | 2 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 7 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 2 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 5 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 0
Dysbiosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Infantile diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 1 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 3 | 8 | 2 | 2 | 2
COVID-19 (Infections and infestations) | 0 | 2 | 5 | 1 | 0 | 11
Nasopharyngitis (Infections and infestations) | 0 | 1 | 2 | 0 | 2 | 4
Bronchitis (Infections and infestations) | 0 | 3 | 2 | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 2 | 1 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Asymptomatic bacteriuria (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Lice infestation (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Otitis media acute (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 0
Suspected COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Vulvovaginitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis rotavirus (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 3 | 1 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Pneumonia klebsiella (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Stoma site infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Bronchitis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Cystitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Enterovirus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Helminthic infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Herpangina (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia moraxella (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia pseudomonal (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Rhinovirus infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Varicella (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Vascular device infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 2 | 1 | 0 | 0 | 0
Acinetobacter infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Enterobacter infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis Escherichia coli (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis adenovirus (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Klebsiella infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0
Klebsiella urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection enterococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 2 | 0 | 3 | 3 | 3 | 8
Procedural headache (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 4 | 13
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 1 | 4
Procedural vomiting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 3
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2
Anaesthetic complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Anaesthetic complication neurological (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Neurological procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Foreign body ingestion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Post procedural fever (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Periorbital haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Post procedural discomfort (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Post procedural swelling (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 4 | 9 | 0 | 1 | 3
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 10 | 1
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Infusion site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Medical device pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Medical device site discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vaccination site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vaccination site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vessel puncture site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Medical device site hypersensitivity (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Medical device site rash (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Respiratory complication associated with device (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 2 | 5 | 0 | 0 | 0
Dairy intolerance (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Underweight (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Lactose intolerance (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Protein deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 2
Joint contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 1 | 1
Short stature (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Tendinous contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Acquired plagiocephaly (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Extremity contracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 1 | 0 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Eczema infantile (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Acne infantile (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0
CSF pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2
Crystal urine present (Investigations) | 0 | 0 | 0 | 0 | 1 | 2
CSF protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Body height below normal (Investigations) | 0 | 0 | 1 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0
Staphylococcus test positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Myocardial necrosis marker increased (Investigations) | 0 | 0 | 3 | 0 | 0 | 0
Bacterial test positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Oxygen saturation decreased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood albumin decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood bicarbonate decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood creatinine decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood phosphorus increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Coronavirus test positive (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1
Leukocyturia (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Peripheral coldness (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cyanosis (Vascular disorders) | 0 | 0 | 2 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vestibular disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 2 | 0 | 0 | 0
Mite allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Milk allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 5 | 0 | 2 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 0 | 0
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Respiratory muscle weakness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Decreased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 3 | 0 | 0 | 0
Hypofibrinogenaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 0 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Secondary thrombocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Myopia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Eye discharge (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 0 | 0 | 2 | 0 | 0 | 0
Cryptorchism (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dysphoria (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2024-06-11): https://cdn.clinicaltrials.gov/large-docs/66/NCT04089566/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-19): https://cdn.clinicaltrials.gov/large-docs/66/NCT04089566/SAP_001.pdf